CLINICAL TRIAL: NCT04776317
Title: A Phase 1 Trial to Evaluate the Safety, Immunogenicity, and Reactogenicity of Heterologous and Homologous Chimpanzee Adenovirus and Self-Amplifying mRNA Prime-Boost Prophylactic Vaccines Against SARS-CoV-2 in Healthy Adults
Brief Title: Chimpanzee Adenovirus and Self-Amplifying mRNA Prime-Boost Prophylactic Vaccines Against SARS-CoV-2 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Gritstone bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0034; 5UM1AI148684-02 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2022-04-20

CONDITIONS: COVID-19
Keywords: Immunogenicity; Prime-Boost; Reactogenicity; Safety; SARS-CoV-2; vaccine
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Stage 1 (Naïve) Group 1 (Experimental): 5 x 10^10 viral particles of ChAdV68-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 30 mcg of SAM-LNP-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 29 in participants from 18 to 60 years of age. N=4
  Interventions: Biological: ChAdV68-S; Biological: SAM-LNP-S; Other: Sodium Chloride, 0.9%
- Stage 1 (Naïve) Group 3A (Experimental): 30 mcg of SAM-LNP-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 30 mcg of SAM-LNP-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 29 in participants from 18 to 60 years of age. N=3
  Interventions: Biological: SAM-LNP-S; Other: Sodium Chloride, 0.9%
- Stage 1 (Naïve) Group 3B (Experimental): 30 mcg SAM-LNP-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 3 mcg of SAM-LNP-S administered through 0.25 mL intramuscular injection in the deltoid muscle on or after Day 85 and no later than Day 130 in participants from 18 to 60 years of age. N=7
  Interventions: Biological: SAM-LNP-S; Other: Sodium Chloride, 0.9%
- Stage 1 (Naïve) Group 4 (Experimental): 10 mcg of SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 3 mcg of SAM-S-TCE administered through 0.25 mL intramuscular injection in the deltoid muscle on or after Day 85 and no later than Day 130 in participants from 18 to 60 years of age. N=3
  Interventions: Biological: SAM-LNP-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 13 (Experimental): 5 x 10^10 viral particles of ChAdV68-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and on or after Day 113 in participants older than 60 years of age. N=7-10
  Interventions: Biological: ChAdV68-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 14 (Experimental): 1 x 10^11 viral particles of ChAdV68-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants older than 60 years of age. N=7-10
  Interventions: Biological: ChAdV68-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 15 (Experimental): 5 x 10^11 viral particles of ChAdV68-S-TCE administered through 1.0 mL intramuscular injection in the deltoid muscle on Day 1 in participants older than 60 years of age. N=7-10
  Interventions: Biological: ChAdV68-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 10A,B (Experimental): 6 mcg of SAM-S-TCE administered through 0.25 mL intramuscular injection in the deltoid muscle on Day 1 in participants older than 60 years of age. N=8-12
  Interventions: Biological: SAM-LNP-S-TCE
- Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 11A,B (Experimental): 10 mcg of SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants older than 60 years of age. N=8-12
  Interventions: Biological: SAM-LNP-S-TCE
- Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 12A,B (Experimental): 10 mcg of SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 10 mcg SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 57 in participants older than 60 years of age. N=8-12
  Interventions: Biological: SAM-LNP-S-TCE
- Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 9 (Experimental): 3 mcg of SAM-S-TCE administered through 0.25 mL intramuscular injection in the deltoid muscle on Day 1 in participants older than 60 years of age. N=8
  Interventions: Biological: SAM-LNP-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 5 (Experimental): 3 mcg of SAM-S-TCE administered through 0.25 mL intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 60 years of age. N=10
  Interventions: Biological: SAM-LNP-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 6 (Experimental): 6 mcg of SAM-S-TCE administered through 0.25 mL intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 60 years of age. N=10
  Interventions: Biological: SAM-LNP-S-TCE; Other: Sodium Chloride, 0.9%
- Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 7A,B (Experimental): 10 mcg of SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants from 18 to 60 years of age. N=8-12
  Interventions: Biological: SAM-LNP-S-TCE
- Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 8A,B (Experimental): 10 mcg of SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 10 mcg of SAM-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 57 in participants from 18 to 60 years of age. N=8-12
  Interventions: Biological: SAM-LNP-S-TCE

INTERVENTIONS:
Biological: ChAdV68-S — Chimpanzee Adenovirus serotype 68 - Spike (ChAdV68-S) is a replication-defective, E1, E3 E4Orf2-4 deleted adenoviral vector based on chimpanzee adenovirus 68 (C68, 68/SAdV-25, originally designated as Pan 9), which belongs to the sub-group E adenovirus family. A single 0.5 mL intramuscular injection will be administered in the deltoid muscle. When possible, the prime vaccine and boost vaccine should be administered in different arms.
  Arms: Stage 1 (Naïve) Group 1
Biological: ChAdV68-S-TCE — Chimpanzee Adenovirus 68 - Spike plus additional SARS-CoV-2 T cell epitopes (ChAdV68-S-TCE) is a replication-defective, E1, E3 E4Orf2-4 deleted adenoviral vector based on chimpanzee adenovirus 68 (C68, 68/SAdV-25, originally designated as Pan 9), which belongs to the sub-group E adenovirus family. A single 0.5- or 1.0-mL (depending on dose level) intramuscular injection will be administered in the deltoid muscle. When possible, the prime vaccine and boost vaccine should be administered in different arms.
  Arms: Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 13; Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 14; Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 15
Biological: SAM-LNP-S — Self-Amplifying mRNA - Lipid Nanoparticles - Spike (SAM-LNP-S) is a SAM vector based on Venezuelan Equine Encephalitis Virus (VEEV). A single 0.25 mL or 0.5 mL (depending on dose level) intramuscular injection will be administered in the deltoid muscle. When possible, the prime vaccine and boost vaccine should be administered in different arms.
  Arms: Stage 1 (Naïve) Group 1; Stage 1 (Naïve) Group 3A; Stage 1 (Naïve) Group 3B
Biological: SAM-LNP-S-TCE — Self-Amplifying mRNA - Lipid Nanoparticles -Spike plus additional SARS-CoV-2 T cell epitopes (SAM-S-TCE) is a SAM vector based on Venezuelan Equine Encephalitis Virus (VEEV). A single 0.25 or 0.5 mL (depending on dose level) intramuscular injection will be administered in the deltoid muscle. When possible, the prime vaccine and boost vaccine should be administered in different arms.
  Arms: Stage 1 (Naïve) Group 4; Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 5; Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 6; Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 7A,B; Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 8A,B; Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 10A,B; Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 11A,B; Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 12A,B; Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 9
Other: Sodium Chloride, 0.9% — The diluent used for this study will be 0.9% Sodium Chloride Injection, USP, and is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection. Each milliliter (mL) contains sodium chloride 9 mg. It contains no bacteriostat, antimicrobial agent or added buffer and is supplied only in single-dose containers to dilute or dissolve drugs for injection. 0.308 mOsmol/mL (calc.). 0.9% Sodium Chloride Injection, USP contains no preservatives.
  Arms: Stage 1 (Naïve) Group 1; Stage 1 (Naïve) Group 3A; Stage 1 (Naïve) Group 3B; Stage 1 (Naïve) Group 4; Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 13; Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 14; Stage 2 (ChAd-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 15; Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 5; Stage 2 (SAM-S-TCE Boosts after EUA/licensed mRNA COVID-19 Vaccines) Group 6; Stage 2 (SAM-S-TCE Boosts after approved/licensed mRNA COVID-19 Vaccines) Group 9

SUMMARY:
This is a multicenter, US-only, phase 1, open-label, dose escalation, non-randomized study of the safety, tolerability, and immunogenicity of investigational ChAd and SAM SARS-CoV-2 vaccines in healthy adult subjects. Homologous and heterologous prime-boost vaccination schedules (Stage 1), as well as boost(s) after receipt of COVID-19 EUA/licensed vaccines (Stage 2) will be examined. Subjects' willingness to receive ChAd vaccines will be assessed and documented at the time of informed consent and considered to determine group assignments. This phase 1 study will enroll 17 Stage 1 and up to 118 Stage 2 subjects. Eligible subjects will be enrolled in different groups based on their age (18-60 years old and >60 years old) and their EUA/licensed COVID-19 vaccination status. A sentinel approach with 72-hour (Stage 1, and Stage 2, Groups 5, 6, 8-10, 12, 13-15) or 7-day observation times (Groups 7 and 11) will be used, before recruiting the remainder of each dose escalation group. Decisions about dose escalation will be determined by the SSC with consultation with the DSMB as needed after all subjects in each group have been observed through Day 8 post first study vaccination. All subjects will be followed through 12 months after their last study vaccination. Vaccinated subjects will be carefully monitored for exposure and infection to SARS-CoV-2 throughout the study. Escalation to the highest dose (10 µg) of SAM-S-TCE in younger subjects will proceed only following safety assessments of the 10 µg dose in older subjects for a period of 28 days post-vaccination. In addition, the dosage of SAM-S-TCE given as a double boost to subjects previously vaccinated with the Johnson & Johnson/Janssen Ad26 COVID-19 EUA/licensed vaccine in Groups 8A, 8B, and 12A, 12B will be determined based on the dose escalation reactogenicity and immunogenicity results in Groups 5-7 and 9-11, respectively. After protocol version 9.0 was implemented, it was decided not to enroll subjects into Groups 7 and 8 because of competing priorities and predicted difficulties enrolling into these two groups.

The primary objectives of this study are 1) To assess the safety and tolerability of different doses of ChAd-S or ChAd-S-TCE, and SAM-S or SAM-S-TCE when administered as prime-boost in healthy naïve adult subjects, 2) To assess the safety and tolerability of different doses of ChAd-S or ChAd-S-TCE, and SAM-S or SAM-S-TCE when administered as first or second boost in healthy adult subjects previously vaccinated with an mRNA or adenoviral-vectored COVID-19 EUA/licensed vaccine.

DETAILED DESCRIPTION:
This is a multicenter, US-only, phase 1, open-label, dose escalation, non-randomized study of the safety, tolerability, and immunogenicity of investigational ChAd and SAM SARS-CoV-2 vaccines in healthy adult subjects. Homologous and heterologous prime-boost vaccination schedules (Stage 1), as well as boost(s) after receipt of COVID-19 EUA/licensed vaccines (Stage 2) will be examined. Subjects' willingness to receive ChAd vaccines will be assessed and documented at the time of informed consent and considered to determine group assignments. This phase 1 study will enroll 17 Stage 1 and up to 118 Stage 2 subjects. Eligible subjects will be enrolled in different groups based on their age (18-60 years old and >60 years old) and their EUA/licensed COVID-19 vaccination status. A sentinel approach with 72-hour (Stage 1, and Stage 2, Groups 5, 6, 8-10, 12, 13-15) or 7-day observation times (Groups 7 and 11) will be used, before recruiting the remainder of each dose escalation group. Decisions about dose escalation will be determined by the SSC with consultation with the DSMB as needed after all subjects in each group have been observed through Day 8 post first study vaccination. All subjects will be followed through 12 months after their last study vaccination. Vaccinated subjects will be carefully monitored for exposure and infection to SARS-CoV-2 throughout the study. Escalation to the highest dose (10 µg) of SAM-S-TCE in younger subjects will proceed only following safety assessments of the 10 µg dose in older subjects for a period of 28 days post-vaccination. In addition, the dosage of SAM-S-TCE given as a double boost to subjects previously vaccinated with the Johnson & Johnson/Janssen Ad26 COVID-19 EUA/licensed vaccine in Groups 8A, 8B, and 12A, 12B will be determined based on the dose escalation reactogenicity and immunogenicity results in Groups 5-7 and 9-11, respectively. After protocol version 9.0 was implemented, it was decided not to enroll subjects into Groups 7 and 8 because of competing priorities and predicted difficulties enrolling into these two groups.

The primary objectives of this study are 1) To assess the safety and tolerability of different doses of ChAd-S or ChAd-S-TCE, and SAM-S or SAM-S-TCE when administered as prime-boost in healthy naïve adult subjects, 2) To assess the safety and tolerability of different doses of ChAd-S or ChAd-S-TCE, and SAM-S or SAM-S-TCE when administered as first or second boost in healthy adult subjects previously vaccinated with an mRNA or adenoviral-vectored COVID-19 EUA/licensed vaccine. The secondary objective of this study is to assess the humoral immunogenicity of ChAd-S or ChAd-S-TCE, and SAM-S or SAM-S-TCE.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to participate in this trial must meet all of the following inclusion criteria:

1. Provide written informed consent prior to initiation of any study procedures
2. Able and willing (in the investigator's opinion) to comply with all study requirements
3. Are men or non-pregnant women aged 18 years or older at enrollment
4. Are in good health*

   *As defined by absence of clinically significant medical conditions defined by the CDC as increasing risk for severe corona virus disease-19 (COVID-19) (see exclusion criteria), or other acute or chronic medical conditions determined by medical history, physical examination (PE), screening laboratory test results, and/or clinical assessment of the investigator that are either listed as exclusion criteria below or in the opinion of the investigator would increase risk for study participation or affect the assessment of the safety of subjects. Chronic medical conditions should be stable for the last 60 days (no hospitalizations, emergency room or urgent care for condition, or invasive medical procedures). Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the participating site PI or appropriate sub- investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes in the 60 days prior to enrollment as well as subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to study vaccination.
5. Agree to refrain from blood donation during the course of the study
6. Plan to remain living in the area for the duration of the study
7. Women of childbearing potential (WOCBP)* must plan to avoid pregnancy for at least 60 days after the last study vaccination and be willing to use an adequate method of contraception** consistently for 30 days prior to first study vaccine and for at least 60 days after the last study vaccine.

   *Not sterilized via bilateral oophorectomy, tubal ligation/salpingectomy, hysterectomy, or successful Essure (R) placement (permanent, non-surgical, non-hormonal sterilization with documented radiological confirmation test at least 90 days after the procedure); still menstruating; or < 1 year has passed since the last menses if menopausal

   **Acceptable methods of birth control include the following: oral contraceptives, injection hormonal contraceptive, implant hormonal contraceptive, hormonal patch, intrauterine device, spermicidal products and barrier methods (such as cervical sponge, diaphragm, or condom with spermicide), abstinence, monogamous with a vasectomized partner, non-male sexual relationship
8. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each study vaccination
9. Vital signs within acceptable ranges:

   * Pulse > 50 and = / < 100 beats per minute
   * Systolic blood pressure (BP) = / < 140 millimeters of mercury (mmHg)
   * Diastolic BP = / < 90 mmHg
   * Oral temperature < 37.8 degrees Celsius (100.0 degrees Fahrenheit)
10. Clinical screening lab evaluations (white blood cell (WBC), hemoglobin (HgB), platelets (PLT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin (T Bili), creatine kinase (CK), serum creatinine (Cr) and prothrombin time (PT)/partial thromboplastin time (PTT)) are within acceptable normal reference ranges at the clinical lab being used* *With the exception that ALT, AST, ALP, and creatinine values that are below the reference range will not be exclusionary as these values below reference range are clinically insignificant. Any other screening lab value outside the reference range that is thought to be clinically insignificant by a site investigator must be discussed with the DMID Medical Officer prior to enrollment.
11. Must agree to genetic testing and storage of samples for secondary research
12. Received at least 2 doses of EUA/licensed mRNA vaccines or at least 1 dose of Ad26 vaccine followed by an mRNA booster, with the last COVID-19 vaccine dose given at least 112 days prior to enrollment (Stage 2 only), as confirmed via CDC vaccination card or other appropriate documentation. Subjects may or may not have been previously infected with SARS-CoV-2.

A subject must meet all of the following criteria to be eligible for leukapheresis:

1. Written informed consent for leukapheresis is provided
2. Weight > / = 110 pounds
3. Screening laboratory evaluations are within acceptable ranges at the site where the leukapheresis procedure will be performed
4. Negative urine or serum pregnancy test at screening and on the day of the leukapheresis procedure for women of childbearing potential
5. Adequate bilateral antecubital venous access
6. No use of blood thinners, aspirin, or nonsteroidal anti-inflammatory drugs (NSAIDs) at least 5 days before the leukapheresis procedure

Exclusion Criteria:

Subjects eligible to participate in this trial must not meet any of the following exclusion criteria:

1. History of prior confirmed (PCR or antigen test positive) COVID-19 less than 112 days prior to enrollment.
2. Positive for anti-nucleoprotein SARS-CoV-2 specific antibody by enzyme-linked immunosorbent assay (ELISA) and had the history of upper respiratory illness (URI) compatible with COVID-19 during the 112 days prior to enrollment (seropositivity without a history of URI during the 112 days prior to enrollment will be considered remotely infected persons eligible for enrollment).
3. Positive nasal swab polymerase chain reaction (PCR) at screening.
4. Body mass index (BMI) > 30 kg/m^2 for Stage 1 participants and BMI > 35 kg/m^2 for Stage 2 participants.
5. Presence of medical comorbidities that would place the subject at increased risk for severe COVID-19*

   *Chronic kidney disease, chronic lung disease (including moderate-to-severe asthma), chronic heart disease (heart failure, coronary artery disease or cardiomyopathies), cerebrovascular disease, diabetes mellitus, chronic liver disease, sickle cell disease
6. Increased risk of occupational exposure to SARS-CoV-2 (healthcare workers and emergency response personnel)*

   *Applies to Stage 1 participants only
7. Prior receipt of an approved/licensed or investigational SARS-CoV-2 vaccine (including under EUA)*, approved or investigational adenovirus-vectored vaccines**, or any other approved or investigational vaccine likely to impact the interpretation of the trial data.

   *Exclusion of prior receipt of EUA/licensed COVID-19 vaccines applies to Stage 1 participants only.

   **With the exception of prior receipt of EUA/licensed Johnson & Johnson/Janssen Ad 26 COVID-19 vaccine which is permitted for Groups 8A, 8B, 12A, and 12B.
8. On current treatment or prevention agents with activity against SARS-CoV-2
9. Current smoking or vaping or history of smoking or vaping in prior year*

   *Applies to Stage 1 participants only
10. Breastfeeding, pregnant, or planning to become pregnant during the course of the study.
11. Participation in another research study involving receipt of an investigational product in the 60 days preceding enrolment or planned use during the study period
12. Receipt or planned receipt of any live, attenuated vaccine within 28 days before or after study vaccination
13. Receipt or planned receipt of any subunit or killed vaccine within 14 days before or after vaccination
14. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of first study vaccination or at any time during the study
15. Any confirmed or suspected immunosuppressive or immunodeficient state, including human immunodeficiency virus (HIV) infection, asplenia, recurrent, severe infections and chronic (more than 14 continuous days) immunosuppressant medication within the past 6 months (inhaled, ophthalmic, and topical steroids are allowed)
16. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including urticaria, respiratory difficulty or abdominal pain (or any immediate allergic reaction of any severity to polysorbate due to potential cross-reactive hypersensitivity with the polyethylene glycol component of the vaccine)
17. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema
18. Any history of anaphylaxis, including but not limited to reaction to vaccination
19. Any history of severe allergic drug reaction
20. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
21. History of serious ongoing, unstable psychiatric condition that in the opinion of the investigator would interfere with study participation
22. Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
23. Bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture or family history of bleeding disorder
24. Recent (within the past 3 months) surgery, immobility, chronic infection, or head trauma that could increase the risks of thrombosis.
25. Suspected or known current alcohol abuse. Suspected or known drug abuse in the 5 years preceding enrollment
26. Seropositive for HIV, hepatitis B surface antigen (HBsAg), or seropositive for hepatitis C virus (antibodies to HCV)
27. Have an acute illness* within 72 hours prior to study vaccination

    *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol
28. History of venous or arterial thrombosis or any known thrombophilic condition including heparin-induced thrombocytopenia (HIT) or family history of thrombosis.
29. History of myocarditis or pericarditis.
30. History of Guillain-Barre Syndrome (GBS).
31. Receiving heparin treatment or on medications associated with increased risk of bleeding or thrombosis.
32. Any other condition that in the opinion of the investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Baylor College of Medicine, Houston, Texas
  - The University of Washington - Virology Research Clinic, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 distinct US-based Infectious Diseases Clinical Research Consortium (IDCRC) sites. The first participant was enrolled on March 25, 2021, and the last participant was enrolled on September 29, 2022.
Pre-assignment Details: Stage 1 studied dose escalation of homologous and heterologous prime-boost vaccination schedules in healthy naïve adult participants. Stage 2 studied booster vaccination(s) in adult participant who previously received Coronavirus Disease 2019 (COVID-19) Emergency Use Authorization (EUA)/licensed vaccines.
Groups:
- Stage 1 (Naïve) Group 1: 5 x 10^10 viral particles of ChAdV68-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 and 30 mcg of SAM-LNP-S administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 29 in participants from 18 to 60 years of age. N=4
  ChAdV68-S: Chimpanzee Adenovirus serotype 68 - Spike (ChAdV68-S) is a replication-defective, E1, E3 E4Orf2-4 deleted adenoviral vector based on chimpanzee adenovirus 68 (C68, 68/SAdV-25, originally designated as Pan 9), which belongs to the sub-group E adenovirus family. A single 0.5 mL intramuscular injection will be administered in the deltoid muscle.
  SAM-LNP-S: Self-Amplifying mRNA - Lipid Nanoparticles - Spike (SAM-LNP-S) is a SAM vector based on Venezuelan Equine Encephalitis Virus (VEEV). A single 0.25 mL or 0.5 mL (depending on dose level) intramuscular injection will be administered in the deltoid muscle. When possible, the prime vaccine and boost vaccine should be administered in different arms.
  Sodium Chloride, 0.9%: The diluent used for this study will be 0.9% Sodium Chloride Injection, USP, and is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection. Each milliliter (mL) contains sodium chloride 9 mg. It contains no bacteriostat, antimicrobial agent or added buffer and is supplied only in single-dose containers to dilute or dissolve drugs for injection. 0.308 mOsmol/mL (calc.). 0.9% Sodium Chloride Injection, USP contains no preservatives.
- Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13: 5 x 10^10 viral particles of ChAdV68-S-TCE administered through 0.5 mL intramuscular injection in the deltoid muscle on Day 1 in participants older than 60 years of age. N=7-10
  ChAdV68-S-TCE: Chimpanzee Adenovirus 68 - Spike plus additional SARS-CoV-2 T cell epitopes (ChAdV68-S-TCE) is a replication-defective, E1, E3 E4Orf2-4 deleted adenoviral vector based on chimpanzee adenovirus 68 (C68, 68/SAdV-25, originally designated as Pan 9), which belongs to the sub-group E adenovirus family. A single 0.5- or 1.0-mL (depending on dose level) intramuscular injection will be administered in the deltoid muscle. When possible, the prime vaccine and boost vaccine should be administered in different arms.
  Sodium Chloride, 0.9%: The diluent used for this study will be 0.9% Sodium Chloride Injection, USP, and is a sterile, nonpyrogenic, isotonic solution of sodium chloride and water for injection. Each milliliter (mL) contains sodium chloride 9 mg. It contains no bacteriostat, antimicrobial agent or added buffer and is supplied only in single-dose containers to dilute or dissolve drugs for injection. 0.308 mOsmol/mL (calc.). 0.9% Sodium Chloride Injection, USP contains no preservatives.
Period: Overall Study
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 7A,B | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 8A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 12A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Started | 4 | 3 | 7 | 3 | 10 | 10 | 0 (Groups 7A,B, 8A,B, and 12A,B were not enrolled because of competing priorities and predicted difficulties enrolling into this group.) | 0 (Groups 7A,B, 8A,B, and 12A,B were not enrolled because of competing priorities and predicted difficulties enrolling into this group.) | 8 | 10 | 10 | 0 (Groups 7A,B, 8A,B, and 12A,B were not enrolled because of competing priorities and predicted difficulties enrolling into this group.) | 7 | 7 | 2
Completed | 4 | 2 | 6 | 3 | 9 | 10 | 0 | 0 | 8 | 10 | 10 | 0 | 7 | 7 | 2
Not Completed | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Groups:
- Stage 1 (Naïve) Group 1: Covid-19 Vaccine and infection Naïve, 18-60years old; received intramuscular (IM) injection of 5 x 10^10 vp ChAd-S followed by 30 µg SAM-S.
- Stage 1 (Naïve) Group 3A: Covid-19 Vaccine and infection Naïve, 18-60years old; received intramuscular (IM) injection of 30 µg SAM-S followed by 30 µg SAM-S.
- Stage 1 (Naïve) Group 3B: Covid-19 Vaccine and infection Naïve, 18-60years old; received intramuscular (IM) injection of 30 µg SAM-S followed by 3 µg SAM-S.
- Stage 1 (Naïve) Group 4: Covid-19 Vaccine and infection Naïve, 18-60years old; received intramuscular (IM) injection of 10 µg SAM-S-TCE followed by 3 µg SAM-S-TCE.
- Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, 18-60 years old, received a single intramuscular (IM) injection of 3 µg SAM-S-TCE.
- Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, 18-60 years old, received a single intramuscular (IM) injection of 6 µg SAM-S-TCE.
- Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, greater than 60 years old, received a single intramuscular (IM) injection of 3 µg SAM-S-TCE.
- Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, greater than 60 years old, received a single intramuscular (IM) injection of 6 µg SAM-S-TCE.
- Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, greater than 60 years old, received a single intramuscular (IM) injection of 10 µg SAM-S-TCE.
- Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, greater than 60 years old, received a single intramuscular (IM) injection of 5x10^10 vp ChAd-S-TCE.
- Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, greater than 60 years old, received a single intramuscular (IM) injection of 1x10^11 vp ChAd-S-TCE.
- Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15: Previously (>/=112 days) dosed with Emergency Use Authorization (EUA)/licensed mRNA vaccine, greater than 60 years old, received a single intramuscular (IM) injection of 5x10^11 vp ChAd-S-TCE.
- Total: Total of all reporting groups
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15 | Total
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.9) | 23.3 (8.4) | 45.4 (11.7) | 29.3 (13.6) | 32.9 (12.6) | 34.0 (8.7) | 63.4 (2.8) | 67.8 (4.7) | 66.0 (4.5) | 69.1 (7.1) | 64.7 (5.3) | 67.5 (3.5) | 51.0 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 0 | 6 | 7 | 5 | 6 | 7 | 5 | 2 | 0 | 42
  Male | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 2 | 5 | 2 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 2 | 7 | 3 | 10 | 9 | 8 | 10 | 10 | 7 | 7 | 2 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 4 | 2 | 7 | 3 | 9 | 9 | 8 | 10 | 10 | 6 | 7 | 2 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Previous COVID-19 Infection [Count of Participants; unit: Participants]
  Previous infection | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 5
  No previous infection | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 8 | 8 | 7 | 6 | 2 | 76
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.23 (3.48) | 21.03 (3.18) | 24.51 (2.11) | 25.57 (3.44) | 23.46 (2.94) | 24.79 (3.05) | 26.03 (4.46) | 24.77 (4.31) | 29.26 (2.69) | 23.33 (4.35) | 26.61 (4.74) | 26.55 (2.47) | 25.00 (3.80)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Any New-onset Chronic Medical Conditions (NOCMCs)
Description: Number of participants that experienced any NOCMCs during the course of the study
Time Frame: Day 1 to study completion through up to 1 year post last dose
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0

2. Primary Outcome: Frequency of Any Potentially Immune-mediated Medical Conditions (PIMMCs)
Description: Number of participants that experienced any PIMMCs during the course of the study
Time Frame: Day 1 to study completion through up to 1 year post last dose
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Frequency of Any Medically Attended Adverse Events (MAAEs)
Description: Number of participants that experienced any MAAEs during the course of the study
Time Frame: Day 1 to study completion through up to 1 year post last dose
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 0 | 1 | 4 | 1 | 4 | 4 | 3 | 3 | 5 | 3 | 1 | 0

4. Primary Outcome: Frequency of Any Laboratory AE
Description: Number of participants that experienced any laboratory AE
Time Frame: Through 7 days post each study vaccination
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 4 | 3 | 7 | 3 | 8 | 8 | 7 | 8 | 10 | 6 | 5 | 0

5. Primary Outcome: Frequency of Any Serious Adverse Events (SAEs)
Description: The number of participants that experience any SAEs from Day 1 to study completion. An AE or suspected adverse reaction is considered serious if, in the view of either the participating site PI or appropriate sub-investigator or the sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 to study completion through up to 1 year post last dose
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Frequency of Systemic Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any systemic solicited AEs through 7 days post any vaccination. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever.
Time Frame: Day 1 through Day 8 for Groups 5, 6, 9, 10, 11, 13, 14 and 15 and through 7 days post any vaccination for Groups 1, 3A, 3b and 4.
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 3 | 5 | 2

7. Primary Outcome: Frequency of Local Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any local solicited AEs through 7 days post any vaccination. Local events include: pain at injection site, erythema, and induration.
Time Frame: as for outcome 6
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 4 | 3 | 7 | 3 | 10 | 8 | 5 | 8 | 9 | 1 | 2 | 1

8. Primary Outcome: Frequency of Any Unsolicited Adverse Events (AEs)
Description: Number of participants who experienced any unsolicited AEs through 28 days post vaccination
Time Frame: Day 1 through Day 29 for Groups 5, 6, 9, 10, 11, 13, 14 and 15 and 28 days post any vaccination for Groups 1, 3A, 3b and 4.
Population: The Safety Analysis population for the study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
Participants | 1 | 2 | 6 | 3 | 10 | 8 | 7 | 7 | 8 | 6 | 5 | 2

9. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against D614G for Groups 1 and 3A
Description: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against D614G. Fold-rise is calculated by dividing post-vaccination titers by the Day 1 Pre-Vaccination 1 titer.
Time Frame: Day 29 Post Vaccination 1, Day 57 Post Vaccination 1 (29 Days Post Vaccination 2), Day 209 Post Vaccination 1 (181 Days Post Vaccination 2), Day 394 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: The mITT population includes all enrolled participants who received at least one dose vaccine and contributed both pre- and at least one post vaccination venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
fold rise
  Day 29 Post Vaccination 1 | 11.90 [3.29 to 43.05] | 4.06 [0.19 to 87.32]
  Day 57 Post Vaccination 1 (29 Days Post Vaccination 2) | 72.48 [26.51 to 198.20] | 2.80 [0.03 to 235.59]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 12.27 [5.47 to 27.52] | 1.57 [0.01 to 477.31]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 573.77 [185.04 to 1779.08] | 66.61 [7.44 to 596.29]

10. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against BA.1 for Groups 1 and 3A
Description: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.1. Fold-rise is calculated by dividing post-vaccination titers by the Day 1 Pre-Vaccination 1 titer.
Time Frame: Day 57 Post Vaccination 1 (29 Days Post Vaccination 2), Day 209 Post Vaccination 1 (181 Days Post Vaccination 2), Day 394 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
fold rise
  Day 57 Post Vaccination 1 (29 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.

11. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against BA.4/5 for Groups 1 and 3A
Description: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.4/5. Fold-rise is calculated by dividing post-vaccination titers by the Day 1 Pre-Vaccination 1 titer.
Time Frame: Day 209 Post Vaccination 1 (181 Days Post Vaccination 2), Day 394 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
fold rise
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.

12. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against D614G for Groups 3B and 4
Description: as for outcome 9
Time Frame: Day 29 Post Vaccination 1, Day 57 Post Vaccination 1, Day 85 Post Vaccination 1, Day 99 Post Vaccination 1, Day 113 Post Vaccination 1, Day 169 Post Vaccination 1, Day 265 Post Vaccination 1, Day 450 Post Vaccination 1
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
fold rise
  Day 29 Post Vaccination 1 | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 9.09 [1.61 to 51.40]
  Day 57 Post Vaccination 1: number analyzed (Participants) | 3 | 3
  Day 57 Post Vaccination 1 | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 1.86 [0.48 to 7.13]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 1.18 [0.77 to 1.80] | 23.98 [5.93 to 96.89]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 1.35 [0.62 to 2.92] | 17.21 [1.50 to 197.75]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 9.98 [1.01 to 98.39]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 258.71 [69.53 to 962.60] | 298.33 [17.42 to 5110.28]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 42.59 [5.68 to 319.58] | 130.72 [1.46 to 11696.94]

13. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against BA.1 for Groups 3B and 4
Description: as for outcome 10
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
fold rise
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 1
  Day 29 Post Vaccination 1 | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post Vaccination 1: number analyzed (Participants) | 0 | 1
  Day 57 Post Vaccination 1 |  | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 1
  Day 85 Post Vaccination 1 | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 1
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 1
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 1.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 2.40 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 1
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 1.93 [0.41 to 9.03] | 4.27 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 1
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 28.25 [1.01 to 787.95] | 42.65 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 1
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 11.46 [0.27 to 492.52] | 13.61 [NA to NA] — 95% CI was not estimable because all values were equal.

14. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against BA.4/5 for Groups 3B and 4
Description: as for outcome 11
Time Frame: Day 169 Post Vac 1 (85 Days Post Vac 2), Day 265 Post Vac 1 (181 Days Post Vac 2), Day 450 Post Vac 1 (366 Days Post Vac 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
fold rise
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab. | NA [NA to NA] — Results were not estimable because pre-vaccination samples were not analyzed for this variant. This variant was not in circulation when the pre-vaccination visit samples were assayed and therefore never tested by the lab.

15. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against D614G for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against D614G. Fold-rise is calculated by dividing post-vaccination titers by the Day 1 Pre-Vaccination titer.
Time Frame: Day 15 Post Vaccination, Day 29 Post Vaccination, Day 85 Post Vaccination, Day 181 Post Vaccination, Day 366 Post Vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
fold rise
  Day 15 Post Vaccination | 3.33 [1.62 to 6.85] | 3.05 [1.20 to 7.80] | 6.64 [2.00 to 22.00] | 1.91 [1.19 to 3.05] | 2.03 [1.01 to 4.07] | 2.15 [0.65 to 7.08] | 1.52 [0.81 to 2.83] | 6.06 [0.00 to 5437456045.79]
  Day 29 Post Vaccination | 5.02 [2.20 to 11.45] | 3.62 [1.26 to 10.38] | 8.07 [2.08 to 31.36] | 2.78 [1.23 to 6.29] | 3.27 [1.45 to 7.38] | 2.90 [0.70 to 11.95] | 2.86 [1.06 to 7.73] | 4.55 [0.00 to 14716523.65]
  Day 85 Post Vaccination | 4.96 [2.10 to 11.69] | 3.38 [1.02 to 11.27] | 10.84 [2.58 to 45.49] | 4.06 [1.19 to 13.85] | 5.79 [2.15 to 15.63] | 11.38 [1.51 to 85.69] | 9.94 [2.41 to 41.02] | 2.76 [0.05 to 154.23]
  Day 181 Post Vaccination | 14.19 [6.03 to 33.40] | 6.75 [1.78 to 25.57] | 18.02 [5.57 to 58.27] | 6.60 [1.31 to 33.17] | 3.27 [1.34 to 8.00] | 13.53 [1.32 to 138.39] | 6.54 [1.42 to 30.08] | 1.88 [0.48 to 7.30]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 30.20 [13.00 to 70.18] | 15.28 [5.05 to 46.21] | 10.01 [3.28 to 30.51] | 4.83 [1.15 to 20.33] | 5.16 [2.02 to 13.18] | 21.98 [2.44 to 198.35] | 2.54 [0.95 to 6.77] | 0.89 [0.00 to 229.48]

16. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against BA.1 for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.1. Fold-rise is calculated by dividing post-vaccination titers by the Day 1 Pre-Vaccination titer.
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
fold rise
  Day 15 Post Vaccination | 4.81 [1.76 to 13.14] | 4.95 [1.64 to 14.94] | 6.49 [2.02 to 20.85] | 1.74 [0.83 to 3.64] | 1.97 [1.07 to 3.63] | 2.01 [0.77 to 5.27] | 1.80 [0.97 to 3.36] | 4.29 [0.00 to 16082568.04]
  Day 29 Post Vaccination | 8.63 [2.72 to 27.36] | 7.14 [1.97 to 25.80] | 9.20 [3.02 to 27.98] | 2.43 [1.09 to 5.41] | 2.88 [1.36 to 6.09] | 2.53 [0.67 to 9.59] | 3.77 [1.55 to 9.13] | 5.26 [0.00 to 189185279.21]
  Day 85 Post Vaccination | 7.76 [2.46 to 24.50] | 7.32 [1.86 to 28.77] | 20.73 [5.74 to 74.87] | 6.54 [1.71 to 25.06] | 4.32 [1.79 to 10.43] | 12.26 [1.00 to 149.82] | 11.77 [3.54 to 39.10] | 3.91 [0.00 to 61879.16]
  Day 181 Post Vaccination | 18.53 [6.50 to 52.83] | 13.39 [2.83 to 63.29] | 56.02 [12.24 to 256.46] | 8.76 [1.53 to 50.19] | 3.35 [1.51 to 7.43] | 15.55 [1.30 to 186.51] | 6.12 [1.52 to 24.60] | 3.12 [0.50 to 19.57]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 86.85 [41.81 to 180.39] | 74.37 [26.44 to 209.18] | 40.58 [10.60 to 155.32] | 11.83 [2.32 to 60.39] | 9.95 [2.73 to 36.30] | 44.10 [6.07 to 320.15] | 4.70 [0.95 to 23.29] | 1.46 [0.00 to 23381.67]

17. Secondary Outcome: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 Against BA.4/5 for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean Fold Rise of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.4/5. Fold-rise is calculated by dividing post-vaccination titers by the Day 1 Pre-Vaccination titer.
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
fold rise
  Day 15 Post Vaccination | 4.32 [1.89 to 9.90] | 3.47 [1.42 to 8.498] | 3.38 [1.03 to 11.09] | 1.01 [0.61 to 1.67] | 2.46 [1.18 to 5.12] | 1.74 [0.73 to 4.17] | 1.85 [1.07 to 3.20] | 4.60 [0.00 to 5401100.08]
  Day 29 Post Vaccination | 6.45 [2.35 to 17.69] | 4.89 [1.65 to 14.54] | 6.11 [1.46 to 25.57] | 1.66 [0.80 to 3.46] | 4.30 [1.89 to 9.79] | 1.82 [0.62 to 5.34] | 3.66 [1.31 to 10.25] | 5.78 [0.00 to 645374779.40]
  Day 85 Post Vaccination | 6.08 [2.37 to 15.55] | 5.43 [1.90 to 15.51] | 5.64 [0.96 to 33.11] | 2.95 [0.74 to 11.76] | 6.58 [2.38 to 18.19] | 11.24 [1.02 to 124.31] | 11.63 [1.96 to 69.03] | 9.14 [3.40 to 24.57]
  Day 181 Post Vaccination | 23.87 [8.73 to 65.27] | 13.56 [2.99 to 61.47] | 12.57 [1.27 to 124.69] | 6.67 [1.16 to 38.38] | 4.43 [1.51 to 12.98] | 21.78 [1.54 to 308.82] | 5.56 [0.72 to 44.13] | 11.12 [0.04 to 3478.54]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 121.91 [40.58 to 366.25] | 108.81 [25.43 to 456.54] | 17.31 [3.99 to 75.02] | 11.53 [1.92 to 69.27] | 25.41 [6.70 to 96.36] | 84.18 [9.28 to 763.81] | 10.54 [1.40 to 79.41] | 6.70 [0.00 to 1391842.10]

18. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against D614G for Groups 1 and 3A
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against D614G
Time Frame: Day 1 Pre-Vaccination 1, Day 29 Post Vaccination 1, Day 57 Post vaccination 1 (29 Days Post Vaccination 2), Day 209 Post Vaccination 1 (181 Days Post Vaccination 2), Day 394 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
titer
  Day 1 Pre-Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 59.4991 [16.4477 to 215.2359] | 20.2886 [0.9428 to 436.6000]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 362.4094 [132.5303 to 991.0228] | 14.0063 [0.1665 to 1177.9649]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 61.3577 [27.3553 to 137.6248] | 7.8418 [0.0258 to 2386.5676]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 2868.8374 [925.2210 to 8895.4181] | 333.0359 [37.2009 to 2981.4568]

19. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against BA.1 for Groups 1 and 3A
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.1
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
titer
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 12.8238 [4.2634 to 38.5724] | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 7.3983 [0.0509 to 1074.6821]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 1611.5218 [162.1484 to 16016.2079] | 28.7301 [8.8988 to 92.7564]

20. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against BA.4/5 for Groups 1 and 3A
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.4/5
Time Frame: Day 209 Post Vaccination 1 (181 Days Post Vaccination 2), Day 394 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
titer
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 16.3926 [3.3992 to 79.0522] | 23.6552 [3.5475 to 157.7338]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 1345.8006 [316.0828 to 5730.0774] | 40.2809 [37.7735 to 42.9548]

21. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against D614G for Groups 3B and 4
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against D614G
Time Frame: Day 1 Pre-Vaccination 1, Day 29 Post Vaccination 1, Day 57 Post Vaccination 1, Day 85 Post Vaccination 1, Day 99 Post Vaccination 1, Day 113 Post Vaccination 1, Day 169 Post Vaccination 1, Day 265 Post Vaccination 1, Day 450 Post Vaccination 1
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
titer
  Day 1 Pre-Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 45.4538 [8.0394 to 256.9892]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 3
  Day 57 Post vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 9.2994 [2.4248 to 35.6642]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 5.8980 [3.8574 to 9.0182] | 119.8892 [29.6697 to 484.4483]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 6.7531 [3.1186 to 14.6237] | 86.0638 [7.4913 to 988.7447]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 49.9195 [5.0654 to 491.9535]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 1293.5494 [347.6573 to 4812.9874] | 1491.6390 [87.0789 to 25551.3913]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 212.9680 [28.3847 to 1597.8817] | 653.5897 [7.3041 to 58484.7192]

22. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against BA.1 for Groups 3B and 4
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.1
Time Frame: as for outcome 21
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
titer
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 4 | 1
  Day 1 Pre-Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 1
  Day 29 Post Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 0 | 1
  Day 57 Post vaccination 1 |  | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 6.6902 [1.9111 to 23.4209]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 6.9420 [3.9689 to 12.1423] | 8.1121 [1.0113 to 65.0699]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 120.5431 [31.7334 to 457.8980] | 95.1328 [16.7198 to 541.2903]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 84.8521 [10.1712 to 707.8690] | 85.4674 [2.2603 to 3231.7721]

23. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against BA.4/5 for Groups 3B and 4
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.4/5
Time Frame: Day 169 Post Vaccination 1 (85 Days Post Vaccination 2), Day 265 Post Vaccination 1 (181 Days Post Vaccination 2), Day 450 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
titer
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 5.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 54.4021 [13.4169 to 220.5873] | 85.2857 [26.9267 to 270.1280]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 25.9869 [2.1788 to 309.9511] | 74.1983 [0.1843 to 29875.2865]

24. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against D614G for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against D614G
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination, Day 29 Post Vaccination, Day 85 Post Vaccination, Day 181 Post Vaccination, Day 366 Post Vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
titer
  Day 1 Pre-Vaccination | 112.8328 [74.9904 to 169.7717] | 405.4138 [163.7296 to 1003.8523] | 102.8466 [43.7058 to 242.0140] | 482.9330 [137.4325 to 1697.0099] | 375.5394 [190.3402 to 740.9358] | 146.8761 [45.1229 to 478.0846] | 430.2308 [92.9329 to 1991.7444] | 1843.1744 [0.3234 to 10504058.3536]
  Day 15 Post Vaccination | 376.1197 [235.0324 to 601.9001] | 1237.9613 [480.9811 to 3186.2961] | 682.4080 [360.8116 to 1290.6475] | 921.5980 [346.0068 to 2454.6999] | 761.2916 [431.8043 to 1342.1935] | 315.1407 [151.7524 to 654.4454] | 652.4332 [191.6513 to 2221.0601] | 11176.4335 [0.0710 to 1758617910.3834]
  Day 29 Post Vaccination | 566.1029 [310.8710 to 1030.8861] | 1468.7289 [530.3009 to 4067.8127] | 829.7727 [390.3204 to 1763.9937] | 1341.1447 [559.6738 to 3213.7810] | 1229.6606 [688.3558 to 2196.6330] | 425.4411 [208.6954 to 867.2936] | 1230.7704 [594.6819 to 2547.2370] | 8381.4354 [14.7590 to 4759715.1788]
  Day 85 Post Vaccination | 559.7445 [298.3456 to 1050.1710] | 1371.6395 [454.2866 to 4141.4273] | 1114.9642 [426.7668 to 2912.9379] | 1963.1115 [1292.6702 to 2981.2762] | 2175.7877 [1014.0073 to 4668.6570] | 1670.9884 [372.7901 to 7490.0121] | 4276.7890 [1271.4749 to 14385.5953] | 5078.3770 [49.8822 to 517016.7435]
  Day 181 Post Vaccination | 1601.5347 [823.4208 to 3114.9483] | 2738.3033 [664.2616 to 11288.1810] | 1853.2904 [545.1221 to 6300.7635] | 3188.0320 [1267.3274 to 8019.6704] | 1229.7755 [675.5304 to 2238.7562] | 1986.5339 [262.9892 to 15005.6244] | 2813.3790 [583.7984 to 13557.9362] | 3462.6712 [2.3614 to 5077595.0850]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 3531.7642 [1394.6079 to 8943.9897] | 6195.9903 [1670.4600 to 22981.8713] | 1029.1579 [368.6714 to 2872.9267] | 2333.8724 [840.6688 to 6479.3176] | 1936.6356 [964.5537 to 3888.3864] | 3228.9682 [746.0332 to 13975.5651] | 1093.8728 [234.7605 to 5096.9292] | 1645.4066 [0.0011 to 2410518823.8906]

25. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against BA.1 for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.1
Time Frame: as for outcome 24
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
titer
  Day 1 Pre-Vaccination | 17.7942 [10.4645 to 30.2577] | 33.4039 [14.5993 to 76.4298] | 11.8710 [7.2241 to 19.5068] | 81.1329 [15.5453 to 423.4417] | 87.9255 [46.7925 to 165.2165] | 48.7041 [18.6670 to 127.0739] | 116.3880 [18.7014 to 724.3415] | 468.5976 [0.4353 to 504394.7664]
  Day 15 Post Vaccination | 85.6574 [35.4915 to 206.7310] | 165.3657 [41.7470 to 655.0362] | 77.0553 [25.3844 to 233.9036] | 141.2683 [33.7834 to 590.7255] | 173.5413 [88.2833 to 341.1356] | 97.9557 [47.8716 to 200.4384] | 209.5990 [42.1687 to 1041.8084] | 2008.1706 [0.5760 to 7001401.5955]
  Day 29 Post Vaccination | 153.6259 [58.3967 to 404.1487] | 238.4406 [50.3259 to 1129.7139] | 109.1945 [40.5282 to 294.2012] | 196.8757 [52.8512 to 733.3804] | 253.2367 [136.9000 to 468.4357] | 123.3706 [47.8388 to 318.1582] | 438.3675 [121.7932 to 1577.8064] | 2467.0800 [0.0739 to 82360112.6459]
  Day 85 Post Vaccination | 138.0929 [52.0824 to 366.1436] | 244.4228 [47.9172 to 1246.7870] | 246.0892 [79.8529 to 758.3938] | 530.9893 [214.1227 to 1316.7668] | 379.9728 [193.7003 to 745.3749] | 596.9179 [78.0512 to 4565.0904] | 1369.4248 [272.2749 to 6887.6128] | 1833.8419 [124.8388 to 26938.5377]
  Day 181 Post Vaccination | 329.7767 [141.6572 to 767.7171] | 447.3343 [102.5193 to 1951.9041] | 665.0024 [139.2378 to 3176.0653] | 711.0995 [250.9232 to 2015.2079] | 294.2032 [145.0665 to 596.6614] | 757.4496 [74.4007 to 7711.3502] | 711.7177 [129.7126 to 3905.1120] | 1459.7959 [8.5217 to 250067.9289]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 1779.4509 [604.7857 to 5235.6489] | 2484.3099 [791.0434 to 7802.0952] | 481.6709 [137.6787 to 1685.1324] | 959.9418 [208.3283 to 4423.2495] | 875.2497 [310.8785 to 2464.1849] | 2147.7815 [591.9922 to 7792.2734] | 546.5955 [40.5298 to 7371.5336] | 685.0752 [0.0000 to 11793589460.228]

26. Secondary Outcome: Geometric Mean of Pseudovirus Neutralization ID50 Against BA.4/5 for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean of Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.4/5
Time Frame: as for outcome 24
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
titer
  Day 1 Pre-Vaccination | 12.5099 [7.2840 to 21.4852] | 23.8982 [11.1513 to 51.2159] | 45.8250 [18.5629 to 113.1251] | 94.0770 [24.5317 to 360.7774] | 38.4049 [15.5880 to 94.6198] | 21.0485 [7.7796 to 56.9487] | 63.8694 [15.6348 to 260.9104] | 124.2137 [1.3374 to 11536.4856]
  Day 15 Post Vaccination | 54.0724 [22.1313 to 132.1128] | 82.9652 [24.0835 to 285.8065] | 154.9099 [69.5129 to 345.2179] | 94.8682 [31.8399 to 282.6637] | 94.5667 [41.9028 to 213.4191] | 36.6182 [10.7558 to 124.6664] | 118.0503 [27.7902 to 501.4678] | 571.0459 [0.0451 to 7223499.3503]
  Day 29 Post Vaccination | 80.7230 [30.7358 to 212.0074] | 116.9255 [28.5017 to 479.6755] | 280.1679 [103.4819 to 758.5292] | 155.9792 [51.1285 to 475.8505] | 165.0762 [80.5052 to 338.4896] | 38.3975 [9.7908 to 150.5874] | 233.6561 [91.3256 to 597.8077] | 717.7161 [0.0006 to 863132368.1932]
  Day 85 Post Vaccination | 76.0077 [29.2176 to 197.7290] | 129.8719 [32.8448 to 513.5278] | 258.4824 [73.2796 to 911.7565] | 277.7532 [110.8690 to 695.8376] | 252.6360 [101.3142 to 629.9702] | 236.6733 [18.6894 to 2997.1096] | 742.6808 [85.4290 to 6456.5250] | 1134.9309 [32.8588 to 39200.0612]
  Day 181 Post Vaccination | 298.6044 [143.5689 to 621.0575] | 324.0669 [58.6172 to 1791.6126] | 575.9687 [91.2214 to 3636.6469] | 627.1003 [173.6712 to 2264.3642] | 170.1065 [67.3139 to 429.8701] | 458.4044 [27.4780 to 7647.3637] | 360.5940 [32.6915 to 3977.4306] | 1380.7990 [0.0475 to 40130153.0367]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 1688.7466 [444.3317 to 6418.3249] | 2600.2491 [446.5774 to 15140.2551] | 793.2778 [316.7655 to 1986.6105] | 1084.8950 [284.6646 to 4134.6809] | 976.0525 [311.5167 to 3058.1940] | 1771.7935 [321.8672 to 9753.2512] | 673.1993 [50.3999 to 8992.0307] | 832.4483 [0.0000 to 16056966235.924]

27. Secondary Outcome: Geometric Mean Titer of RBD IgG as Measured by ELISA for Groups 1 and 3A
Description: Geometric Mean of RBD titer
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
titer
  Day 1 Pre-Vaccination 1 | 1.4663 [0.7258 to 2.9623] | 1.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 4.0128 [3.1921 to 5.0445] | 1.3351 [0.3850 to 4.6304]
  Day 57 Post Vaccination 1 (29 Days Post Vaccination 2) | 5.2779 [4.1399 to 6.7286] | 2.3206 [1.8668 to 2.8847]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 4.3994 [3.3972 to 5.6972] | 1.5100 [0.0080 to 283.7685]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 6.5014 [6.1134 to 6.9140] | 5.8002 [2.3386 to 14.3857]

28. Secondary Outcome: Geometric Mean Titer of RBD IgG as Measured by ELISA for Groups 3B and 4
Description: Geometric Mean of RBD titer
Time Frame: as for outcome 21
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
titer
  Day 1 Pre-Vaccination 1 | 1.3894 [0.9495 to 2.0331] | 1.8018 [0.5013 to 6.4767]
  Day 29 Post Vaccination 1 | 1.4036 [0.9473 to 2.0797] | 3.4419 [1.9292 to 6.1409]
  Day 57 Post Vaccination 1: number analyzed (Participants) | 3 | 3
  Day 57 Post Vaccination 1 | 1.0000 [NA to NA] — 95% CI was not estimable because all values were equal. | 3.3980 [1.8922 to 6.1019]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 1.5076 [0.9402 to 2.4175] | 3.5077 [2.2207 to 5.5406]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 1.7037 [1.0986 to 2.6421] | 4.3799 [2.5683 to 7.4694]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 1.5587 [0.9254 to 2.6253] | 4.1463 [2.8173 to 6.1023]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 1.3002 [0.8457 to 1.9989] | 3.9733 [2.8684 to 5.5037]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 5.8158 [5.2752 to 6.4118] | 5.2318 [3.5862 to 7.6325]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 4.7615 [3.7723 to 6.0101] | 5.2214 [2.9214 to 9.3321]

29. Secondary Outcome: Geometric Mean in Titer of RBD IgG as Measured by ELISA for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean of RBD titer
Time Frame: as for outcome 24
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
titer
  Day 1 Pre-Vaccination | 5.5864 [5.2027 to 5.9984] | 6.1054 [5.6569 to 6.5895] | 4.8833 [4.4472 to 5.3623] | 5.2627 [4.6084 to 6.0099] | 5.1098 [4.5935 to 5.6842] | 4.3709 [3.9083 to 4.8882] | 4.7219 [3.6673 to 6.0797] | 5.1950 [5.0078 to 5.3891]
  Day 15 Post Vaccination | 6.1134 [5.8874 to 6.3480] | 6.3735 [6.0264 to 6.7406] | 5.4103 [4.9309 to 5.9362] | 5.5201 [5.0123 to 6.0792] | 5.2454 [4.8127 to 5.7169] | 4.6996 [4.3467 to 5.0811] | 4.8502 [4.1286 to 5.6979] | 6.3734 [2.9596 to 13.7249]
  Day 29 Post Vaccination | 6.1962 [5.7981 to 6.6217] | 6.2725 [5.9372 to 6.6266] | 5.5427 [5.1023 to 6.0211] | 5.2341 [4.8568 to 5.6407] | 5.4238 [5.1794 to 5.6798] | 4.7917 [4.4116 to 5.2046] | 5.1222 [4.4543 to 5.8903] | 6.1749 [5.7458 to 6.6360]
  Day 85 Post Vaccination | 5.9271 [5.6065 to 6.2659] | 6.2709 [5.8290 to 6.7462] | 5.5019 [5.0364 to 6.0103] | 5.3951 [4.9673 to 5.8598] | 5.6756 [5.1714 to 6.2289] | 5.4978 [4.8782 to 6.1960] | 5.7671 [5.1604 to 6.4451] | 6.5832 [3.6902 to 11.7441]
  Day 181 Post Vaccination | 6.1082 [5.7059 to 6.5388] | 6.3086 [5.8666 to 6.7838] | 5.4872 [4.8885 to 6.1593] | 5.5874 [5.1392 to 6.0747] | 5.4714 [4.9852 to 6.0050] | 5.5399 [4.7833 to 6.4160] | 5.6336 [4.8726 to 6.5134] | 6.2200 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 5.6975 [5.2935 to 6.1324] | 5.8714 [5.3733 to 6.4157] | 5.8233 [5.3127 to 6.3829] | 5.9260 [5.4429 to 6.4519] | 5.8235 [5.2837 to 6.4185] | 6.0125 [5.4342 to 6.6523] | 5.3922 [4.4939 to 6.4702] | 5.5803 [2.6334 to 11.8249]

30. Secondary Outcome: Geometric Mean Titer of S-2P IgG as Measured by ELISA for Groups 1 and 3A
Description: Geometric Mean of S-2P titer
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
titer
  Day 1 Pre-Vaccination 1 | 1.8212 [0.9598 to 3.4558] | 1.0000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 4.0618 [3.4563 to 4.7734] | 1.9543 [0.4462 to 8.5590]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 4.7630 [3.8490 to 5.8940] | 2.6772 [1.4588 to 4.9135]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 3.5022 [3.0395 to 4.0353] | 1.6279 [0.0033 to 795.3299]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 5.6119 [4.8366 to 6.5116] | 4.6257 [2.6709 to 8.0111]

31. Secondary Outcome: Geometric Mean Titer of S-2P IgG as Measured by ELISA for Groups 3B and 4
Description: Geometric Mean of S-2P titer
Time Frame: as for outcome 21
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
titer
  Day 1 Pre-Vaccination 1 | 1.2425 [0.8811 to 1.7521] | 1.3426 [0.3780 to 4.7688]
  Day 29 Post Vaccination 1 | 2.2027 [1.5276 to 3.1764] | 3.3798 [2.4180 to 4.7244]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 3
  Day 57 Post vaccination 1 | 2.3213 [0.3589 to 15.0141] | 3.3500 [2.4830 to 4.5198]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 2.0479 [1.1017 to 3.8068] | 3.2201 [2.6540 to 3.9070]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 2.3037 [1.3810 to 3.8429] | 4.0985 [2.5970 to 6.4679]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 2.0917 [1.0950 to 3.9956] | 3.9677 [2.8054 to 5.6116]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 2.6905 [2.0117 to 3.5983] | 3.5196 [2.5478 to 4.8622]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 5.1576 [4.5793 to 5.8088] | 4.7234 [3.3074 to 6.7455]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 4.5632 [3.7534 to 5.5478] | 4.8462 [2.7734 to 8.4683]

32. Secondary Outcome: Geometric Mean in Titer of S-2P IgG as Measured by ELISA for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Geometric Mean of S-2P titer
Time Frame: as for outcome 24
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
titer
  Day 1 Pre-Vaccination | 5.2906 [5.0215 to 5.5741] | 5.6841 [5.2149 to 6.1955] | 4.5982 [4.2377 to 4.9893] | 5.2196 [4.6659 to 5.8390] | 5.1658 [4.7844 to 5.5778] | 4.5890 [3.9383 to 5.3472] | 5.3462 [4.6020 to 6.2108] | 5.1096 [2.8489 to 9.1641]
  Day 15 Post Vaccination | 5.7415 [5.5118 to 5.9807] | 6.0642 [5.6893 to 6.4639] | 5.0168 [4.6097 to 5.4600] | 5.2691 [4.8097 to 5.7724] | 5.5084 [5.1758 to 5.8623] | 5.0731 [4.6581 to 5.5252] | 5.3743 [4.6002 to 6.2786] | 6.1184 [3.3860 to 11.0557]
  Day 29 Post Vaccination | 6.0318 [5.6884 to 6.3960] | 6.0754 [5.6760 to 6.5028] | 5.1947 [4.6974 to 5.7447] | 5.5926 [5.1392 to 6.0859] | 5.6533 [5.4356 to 5.8797] | 5.0920 [4.5783 to 5.6633] | 5.6380 [5.0530 to 6.2907] | 5.5236 [4.1434 to 7.3636]
  Day 85 Post Vaccination | 5.7937 [5.5268 to 6.0734] | 6.0462 [5.5754 to 6.5569] | 4.8845 [4.4528 to 5.3580] | 5.1933 [4.8645 to 5.5444] | 5.8548 [5.4504 to 6.2892] | 5.4640 [4.8358 to 6.1737] | 5.8416 [5.1800 to 6.5878] | 6.4489 [5.0911 to 8.1689]
  Day 181 Post Vaccination | 5.5115 [5.0201 to 6.0510] | 5.5887 [4.9609 to 6.2961] | 4.7663 [4.3033 to 5.2790] | 5.2681 [4.8152 to 5.7635] | 5.5167 [5.1231 to 5.9405] | 5.5953 [4.8132 to 6.5044] | 5.6251 [4.8903 to 6.4703] | 5.7356 [0.7961 to 41.3242]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 5.1647 [4.7379 to 5.6300] | 5.5361 [4.9747 to 6.1608] | 4.8448 [4.5241 to 5.1882] | 5.3569 [4.8486 to 5.9184] | 5.3687 [4.9860 to 5.7809] | 5.3688 [4.6880 to 6.1484] | 5.1322 [4.4562 to 5.9108] | 5.0425 [1.7521 to 14.5125]

33. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against D614G S-2P for Groups 1 and 3A
Description: Percent of Participants Who Seroconverted, defined as a 4-fold change in Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against D614G S-2P
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percentage of participants
  Day 29 Post Vaccination 1 | 100 [40 to 100] | 67 [9 to 99]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 100 [40 to 100] | 33 [1 to 91]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 100 [40 to 100] | 50 [1 to 99]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 100 [40 to 100] | 100 [16 to 100]

34. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against BA.1 S-2P for Groups 1 and 3A
Description: Percent of Participants Who Seroconverted, defined as a 4-fold change in Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.1 S-2P
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percentage of participants
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 75 [19 to 99] | 0 [0 to 71]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 0 [0 to 60] | 50 [1 to 99]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 100 [40 to 100] | 100 [16 to 100]

35. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against BA.4/5 S-2P for Groups 1 and 3A
Description: Percent of Participants Who Seroconverted, defined as a 4-fold change in Pseudovirus Neutralization ID50 (50% Inhibitory Dilution) against BA.4/5 S-2P
Time Frame: Day 209 Post Vaccination 1 (181 Days Post Vaccination 2), Day 394 Post Vaccination 1 (366 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percentage of participants
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 75 [19 to 99] | 100 [16 to 100]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 100 [40 to 100] | 100 [16 to 100]

36. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against D614G S-2P for Groups 3B and 4
Description: as for outcome 33
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of participants
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 100 [29 to 100]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 3
  Day 57 Post vaccination 1 | 0 [0 to 71] | 67 [9 to 99]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 17 [1 to 64] | 100 [29 to 100]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 17 [1 to 64] | 100 [29 to 100]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 0 [0 to 46] | 100 [29 to 100]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 100 [48 to 100] | 100 [29 to 100]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 100 [48 to 100] | 100 [29 to 100]

37. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against BA.1 S-2P for Groups 3B and 4
Description: Percent of Participants Who Seroconverted, defined as a 4-fold change in Pseudovirus Neutralization ID50 (50% Inhibitory Dilution), against BA.1 S-2P
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of participants
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 1
  Day 29 Post Vaccination 1 | 0 [0 to 60] | 0 [0 to 98]
  Day 57 Post vaccination 1: number analyzed (Participants) | 0 | 1
  Day 57 Post vaccination 1 |  | 0 [0 to 98]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 0 [0 to 46] | 33 [1 to 91]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 33 [4 to 78] | 33 [1 to 91]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 100 [48 to 100] | 100 [29 to 100]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 100 [48 to 100] | 100 [29 to 100]

38. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against BA.4/5 S-2P for Groups 3B and 4
Description: Percent of Participants Who Seroconverted, defined as a 4-fold change in Pseudovirus Neutralization ID50 (50% Inhibitory Dilution), against BA.4/5 S-2P
Time Frame: as for outcome 23
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of participants
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 100 [48 to 100] | 100 [29 to 100]
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 450 Post Vaccination 1 (366 Days Post Vaccination 2) | 60 [15 to 95] | 100 [29 to 100]

39. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against D614G S-2P for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Percent of Participants Who Seroconverted, defined as a 4-fold change in Pseudovirus Neutralization ID50 (50% Inhibitory Dilution), against D614G S-2P
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of participants
  Day 15 Post Vaccination | 100 [69 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 29 Post Vaccination | 100 [69 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 85 Post Vaccination | 100 [69 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 181 Post Vaccination | 100 [69 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 100 [66 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]

40. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against BA.1 S-2P for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 37
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of participants
  Day 15 Post Vaccination | 100 [69 to 100] | 90 [55 to 99] | 100 [63 to 100] | 90 [55 to 99] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 29 Post Vaccination | 100 [69 to 100] | 90 [55 to 99] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 85 Post Vaccination | 100 [69 to 100] | 90 [55 to 99] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 181 Post Vaccination | 100 [69 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 100 [66 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 86 [42 to 99] | 100 [16 to 100]

41. Secondary Outcome: Percent of Participants Who Seroconverted Based on Pseudovirus Neutralization ID50 Against BA.4/5 S-2P for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 38
Time Frame: as for outcome 15
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of participants
  Day 15 Post Vaccination | 90 [55 to 99] | 90 [55 to 99] | 100 [63 to 100] | 90 [55 to 99] | 100 [69 to 100] | 86 [42 to 99] | 100 [59 to 100] | 100 [16 to 100]
  Day 29 Post Vaccination | 90 [55 to 99] | 90 [55 to 99] | 100 [63 to 100] | 90 [55 to 99] | 100 [69 to 100] | 86 [42 to 99] | 100 [59 to 100] | 100 [16 to 100]
  Day 85 Post Vaccination | 90 [55 to 99] | 90 [55 to 99] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 181 Post Vaccination | 100 [69 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]
  Day 366 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 10 | 10 | 7 | 7 | 2
  Day 366 Post Vaccination | 100 [66 to 100] | 100 [69 to 100] | 100 [63 to 100] | 100 [69 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [59 to 100] | 100 [16 to 100]

42. Secondary Outcome: Mean Percent of CD4+ T Cells With Any COV2 S Stimulation Expressing IFNg and/or IL-2 for Groups 1 and 3A
Description: Mean Percent of CD4+ T Cells with Any COV2 S stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 29 Post Vaccination 1, Day 57 Post vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 4 | 2
  Day 1 Pre-Vaccination | 0.033 [-0.031 to 0.098] | 0.040 [-0.109 to 0.190]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 2
  Day 29 Post Vaccination 1 | 0.294 [-0.098 to 0.687] | 0.078 [-0.896 to 1.051]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 0.216 [0.006 to 0.427] | 0.090 [-0.819 to 1.000]

43. Secondary Outcome: Mean Percent of CD4+ T Cells With Any COV2 S Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 1 and 3A
Description: Mean Percent of CD4+ T Cells with Any COV2 S stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: Day 1 Pre-Vaccination, Day 29 Post Vaccination 1, Day 57 Post vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 4 | 2
  Day 1 Pre-Vaccination | 0.003 [-0.004 to 0.011] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 2
  Day 29 Post Vaccination 1 | 0.024 [-0.023 to 0.071] | 0.004 [-0.035 to 0.043]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 0.013 [-0.026 to 0.053] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.

44. Secondary Outcome: Mean Percent of CD4+ T Cells With Any COV2 S Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with Any COV2 S stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 29 Post Vaccination 1, Day 85 Post Vaccination 1, Day 99 Post vaccination 1 (15 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.007 [0.002 to 0.012] | 0.012 [-0.034 to 0.057]
  Day 29 Post Vaccination 1 | 0.017 [-0.003 to 0.037] | 0.026 [-0.074 to 0.126]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.011 [-0.007 to 0.029] | 0.017 [-0.005 to 0.040]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.028 [0.005 to 0.052] | 0.016 [-0.007 to 0.039]

45. Secondary Outcome: Mean Percent of CD4+ T Cells With Any COV2 S Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with Any COV2 S stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.002 [-0.001 to 0.005] | 0.015 [-0.046 to 0.077]
  Day 29 Post Vaccination 1 | 0.001 [0.001 to 0.002] | 0.019 [-0.059 to 0.097]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.002 [-0.001 to 0.005] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.003 [0.000 to 0.005] | 0.004 [-0.010 to 0.019]

46. Secondary Outcome: Mean Percent of CD4+ T Cells With Any TCE Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with Any TCE stimulation expressing IFNg and/or IL-2
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.003 [0.001 to 0.005] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 0.002 [-0.001 to 0.005] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.001 [0.001 to 0.001] | 0.003 [-0.005 to 0.011]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.003 [-0.006 to 0.011]

47. Secondary Outcome: Mean Percent of CD4+ T Cells With Any TCE Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with Any TCE stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.007 [-0.019 to 0.033]
  Day 29 Post Vaccination 1 | 0.002 [-0.000 to 0.004] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.006 [-0.002 to 0.013] | 0.001 [0.000 to 0.003]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.004 [-0.001 to 0.009] | 0.005 [-0.013 to 0.024]

48. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Mem Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with G-Mem stimulation expressing IFNg and/or IL-2
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.004 [0.001 to 0.007] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 0.002 [0.000 to 0.005] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.001 [0.000 to 0.003] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.002 [-0.000 to 0.004] | 0.001 [0.001 to 0.001]

49. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Mem Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with G-Mem stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.002 [0.000 to 0.003] | 0.002 [-0.001 to 0.004]
  Day 29 Post Vaccination 1 | 0.001 [0.000 to 0.003] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.002 [-0.001 to 0.006] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.

50. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Nuc Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with G-Nuc stimulation expressing IFNg and/or IL-2
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 0.001 [0.001 to 0.002] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.004 [-0.010 to 0.018]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.005 [-0.011 to 0.020]

51. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Nuc Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with G-Nuc stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.003 [-0.005 to 0.011]
  Day 29 Post Vaccination 1 | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.001 [-0.000 to 0.003]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.003 [-0.001 to 0.007] | 0.001 [-0.000 to 0.003]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.001 [0.000 to 0.003] | 0.004 [-0.010 to 0.019]

52. Secondary Outcome: Mean Percent of CD4+ T Cells With G-ORFa Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with G-ORFa stimulation expressing IFNg and/or IL-2
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.002 [0.000 to 0.004] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 0.001 [0.001 to 0.002] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.001 [0.001 to 0.001] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.

53. Secondary Outcome: Mean Percent of CD4+ T Cells With G-ORFa Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Mean Percent of CD4+ T Cells with G-ORFa stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.004 [-0.009 to 0.017]
  Day 29 Post Vaccination 1 | 0.004 [-0.000 to 0.008] | 0.006 [-0.016 to 0.028]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0.005 [-0.002 to 0.011] | 0.002 [-0.003 to 0.008]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0.004 [-0.003 to 0.012] | 0.003 [-0.007 to 0.014]

54. Secondary Outcome: Mean Percent of CD4+ T Cells With Any COV2 S Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with Any COV2 S stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.284 [0.028 to 0.540] | 0.315 [0.032 to 0.598] | 0.182 [0.046 to 0.318] | 0.099 [0.018 to 0.180] | 0.237 [0.091 to 0.383] | 0.166 [0.060 to 0.272] | 0.149 [-0.005 to 0.304] | 0.103 [-0.563 to 0.768]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.192 [0.108 to 0.276] | 0.316 [0.084 to 0.547] | 0.225 [0.098 to 0.353] | 0.111 [0.029 to 0.193] | 0.252 [0.139 to 0.365] | 0.172 [0.082 to 0.262] | 0.228 [0.014 to 0.443] | 0.223 [-1.995 to 2.442]

55. Secondary Outcome: Mean Percent of CD4+ T Cells With Any COV2 S Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with Any COV2 S stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.018 [-0.018 to 0.053] | 0.005 [0.000 to 0.009] | 0.018 [-0.002 to 0.037] | 0.006 [0.001 to 0.010] | 0.015 [-0.003 to 0.033] | 0.007 [-0.006 to 0.020] | 0.004 [-0.001 to 0.009] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.003 [-0.001 to 0.008] | 0.008 [-0.000 to 0.016] | 0.004 [0.001 to 0.008] | 0.004 [-0.000 to 0.008] | 0.015 [0.000 to 0.029] | 0.004 [-0.003 to 0.011] | 0.012 [-0.001 to 0.025] | 0.003 [-0.019 to 0.024]

56. Secondary Outcome: Mean Percent of CD4+ T Cells With Any TCE Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with Any TCE stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.016 [-0.003 to 0.034] | 0.011 [-0.001 to 0.024] | 0.002 [-0.000 to 0.005] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.010 [-0.009 to 0.028] | 0.007 [-0.006 to 0.019] | 0.002 [-0.000 to 0.005] | 0.003 [-0.019 to 0.025]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.019 [-0.005 to 0.043] | 0.015 [0.000 to 0.030] | 0.022 [-0.023 to 0.067] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.014 [-0.004 to 0.033] | 0.007 [-0.001 to 0.014] | 0.011 [-0.005 to 0.027] | 0.006 [-0.016 to 0.028]

57. Secondary Outcome: Mean Percent of CD4+ T Cells With Any TCE Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with Any TCE stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.004 [-0.000 to 0.008] | 0.003 [-0.000 to 0.006] | 0.036 [-0.024 to 0.097] | 0.005 [-0.001 to 0.011] | 0.005 [-0.002 to 0.012] | 0.012 [-0.001 to 0.025] | 0.008 [0.000 to 0.016] | 0.011 [-0.006 to 0.029]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.001 [0.001 to 0.002] | 0.004 [0.000 to 0.007] | 0.006 [-0.002 to 0.013] | 0.003 [-0.001 to 0.007] | 0.005 [-0.001 to 0.011] | 0.002 [-0.001 to 0.005] | 0.004 [-0.001 to 0.009] | 0.001 [-0.005 to 0.008]

58. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Mem Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with G-Mem stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.011 [0.001 to 0.021] | 0.011 [0.003 to 0.019] | 0.001 [0.000 to 0.002] | 0.002 [-0.000 to 0.004] | 0.002 [-0.001 to 0.005] | 0.001 [0.001 to 0.002] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.001 [-0.003 to 0.006]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.014 [-0.004 to 0.033] | 0.011 [0.003 to 0.019] | 0.002 [0.001 to 0.002] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.003 [0.000 to 0.006] | 0.003 [-0.001 to 0.006] | 0.005 [0.000 to 0.009] | 0.002 [-0.014 to 0.019]

59. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Mem Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with G-Mem stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.003 [0.001 to 0.005] | 0.001 [0.001 to 0.002] | 0.008 [-0.006 to 0.023] | 0.002 [0.000 to 0.004] | 0.003 [-0.000 to 0.005] | 0.002 [0.000 to 0.003] | 0.002 [0.000 to 0.005] | 0.002 [-0.014 to 0.019]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.002 [-0.000 to 0.004] | 0.003 [0.000 to 0.005] | 0.003 [-0.001 to 0.006] | 0.002 [0.001 to 0.003] | 0.001 [0.001 to 0.002] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.002 [0.000 to 0.003] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.

60. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Nuc Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with G-Nuc stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.003 [-0.000 to 0.007] | 0.001 [0.001 to 0.002] | 0.001 [0.000 to 0.003] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.007 [-0.002 to 0.016] | 0.005 [-0.001 to 0.010] | 0.008 [-0.007 to 0.023] | 0.004 [-0.034 to 0.042]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.002 [-0.000 to 0.004] | 0.002 [0.001 to 0.003] | 0.019 [-0.021 to 0.058] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.008 [-0.001 to 0.017] | 0.008 [-0.004 to 0.019] | 0.010 [-0.012 to 0.033] | 0.003 [-0.018 to 0.024]

61. Secondary Outcome: Mean Percent of CD4+ T Cells With G-Nuc Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with G-Nuc stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.001 [0.001 to 0.002] | 0.006 [-0.003 to 0.015] | 0.012 [-0.009 to 0.034] | 0.002 [0.000 to 0.004] | 0.004 [-0.002 to 0.010] | 0.005 [-0.001 to 0.012] | 0.002 [0.001 to 0.003] | 0.011 [-0.081 to 0.103]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.001 [0.001 to 0.001] | 0.001 [0.001 to 0.002] | 0.005 [-0.003 to 0.012] | 0.002 [0.000 to 0.003] | 0.002 [0.001 to 0.003] | 0.003 [-0.001 to 0.007] | 0.002 [-0.000 to 0.005] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.

62. Secondary Outcome: Mean Percent of CD4+ T Cells With G-ORFa Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with G-ORFa stimulation expressing IFNg and/or IL-2
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 9 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.006 [-0.002 to 0.014] | 0.005 [-0.002 to 0.012] | 0.002 [-0.000 to 0.004] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.004 [-0.003 to 0.011] | 0.003 [-0.002 to 0.009] | 0.003 [-0.001 to 0.008] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.004 [-0.002 to 0.011] | 0.009 [-0.001 to 0.019] | 0.007 [-0.005 to 0.019] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.006 [-0.002 to 0.014] | 0.001 [0.001 to 0.002] | 0.003 [0.001 to 0.006] | 0.005 [-0.044 to 0.055]

63. Secondary Outcome: Mean Percent of CD4+ T Cells With G-ORFa Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: Mean Percent of CD4+ T Cells with G-ORFa stimulation expressing IL-4 or IL-5 or IL-13 and CD154
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: percentage of CD4+ T Cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percentage of CD4+ T Cells
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 9 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0.002 [0.000 to 0.004] | 0.002 [0.000 to 0.003] | 0.020 [-0.004 to 0.044] | 0.003 [-0.000 to 0.006] | 0.001 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.009 [0.001 to 0.017] | 0.009 [-0.003 to 0.021] | 0.003 [-0.023 to 0.029]
  Day 15 Post Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post Vaccination | 0.001 [0.001 to 0.002] | 0.002 [-0.000 to 0.004] | 0.001 [0.001 to 0.002] | 0.002 [0.000 to 0.004] | 0.005 [-0.001 to 0.010] | 0.005 [-0.004 to 0.015] | 0.004 [-0.002 to 0.010] | 0.006 [-0.061 to 0.074]

64. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any COV2 S Stimulation Expressing IFNg and/or IL-2 for Groups 1 and 3A
Description: Percent of Responders: CD4+ T Cells with Any COV2 S stimulation expressing IFNg and/or IL-2.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-values using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: Day 1 Pre-Vaccination, Day 29 Post Vaccination 1, Day 57 Post vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 4 | 2
  Day 1 Pre-Vaccination | 25 [1 to 81] | 50 [1 to 99]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 2
  Day 29 Post Vaccination 1 | 75 [19 to 99] | 50 [1 to 99]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 75 [19 to 99] | 50 [1 to 99]

65. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any COV2 S Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 1 and 3A
Description: Percent of Responders: CD4+ T Cells with Any COV2 S stimulation expressing IL-4 or IL-5 or IL-13 and CD154
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-vals using the Bonferroni-Holm adjustment method. If the adjusted p-val for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: Day 1 Pre-Vaccination, Day 29 Post Vaccination 1, Day 57 Post vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 4 | 2
  Day 1 Pre-Vaccination | 0 [0 to 60] | 0 [0 to 84]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 4 | 2
  Day 29 Post Vaccination 1 | 0 [0 to 60] | 0 [0 to 84]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 25 [1 to 81] | 0 [0 to 84]

66. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any COV2 S Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: as for outcome 64
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

67. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any COV2 S Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with Any COV2 S stimulation expressing IL-4 or IL-5 or IL-13 and CD154.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-vals using the Bonferroni-Holm adjustment method. If the adjusted p-val for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 1 [1 to 91]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

68. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any TCE Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with Any TCE stimulation expressing IFNg and/or IL-2.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-values using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

69. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any TCE Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with Any TCE stimulation expressing IL-4 or IL-5 or IL-13 and CD154.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-vals using the Bonferroni-Holm adjustment method. If the adjusted p-val for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

70. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Mem Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with G-Mem stimulation expressing IFNg and/or IL-2.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-values using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

71. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Mem Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with G-Mem stimulation expressing IL-4 or IL-5 or IL-13 and CD154.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-vals using the Bonferroni-Holm adjustment method. If the adjusted p-val for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

72. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Nuc Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with G-Nuc stimulation expressing IFNg and/or IL-2.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-values using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

73. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Nuc Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with G-Nuc stimulation expressing IL-4 or IL-5 or IL-13 and CD154.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-vals using the Bonferroni-Holm adjustment method. If the adjusted p-val for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

74. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-ORFa Stimulation Expressing IFNg and/or IL-2 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with G-ORFa stimulation expressing IFNg and/or IL-2.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-values using the Bonferroni-Holm adjustment method. If the adjusted p-value for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

75. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-ORFa Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 3B and 4
Description: Percent of Responders: CD4+ T Cells with G-ORFa stimulation expressing IL-4 or IL-5 or IL-13 and CD154.
  To assess positivity for a peptide pool within a T cell subset, a two-by-two contingency table was constructed comparing the stimulated and negative control data. The four entries in each table were the number of cells positive for the cytokine of interest and the number of cells negative for the cytokine, for both the stimulated and the negative control data. A one-sided Fisher's exact test was applied to the table, testing whether the number of cytokine-producing cells for the stimulated data was equal to that for the negative control data. Since multiple individual tests (for each peptide pool) were conducted simultaneously, a multiplicity adjustment was made to the individual peptide pool p-vals using the Bonferroni-Holm adjustment method. If the adjusted p-val for a peptide pool was =0.00001, the response to the peptide pool for the T cell subset was considered positive.
Time Frame: as for outcome 44
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
percent of responders
  Day 1 Pre-Vaccination | 0 [0 to 41] | 0 [0 to 71]
  Day 29 Post Vaccination 1 | 0 [0 to 41] | 0 [0 to 71]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 85 Post Vaccination 1 | 0 [0 to 46] | 0 [0 to 71]
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 99 Post vaccination 1 (15 Days Post Vaccination 2) | 0 [0 to 46] | 0 [0 to 71]

76. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any COV2 S Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 64
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 70 [35 to 93] | 80 [44 to 97] | 63 [24 to 91] | 38 [9 to 76] | 70 [35 to 93] | 67 [22 to 96] | 57 [18 to 90] | 50 [1 to 99]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 89 [52 to 99] | 80 [44 to 97] | 100 [63 to 100] | 56 [21 to 86] | 80 [44 to 97] | 67 [22 to 96] | 86 [42 to 99] | 50 [1 to 99]

77. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any COV2 S Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 67
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 10 [1 to 45] | 0 [0 to 31] | 13 [1 to 53] | 0 [0 to 37] | 20 [3 to 56] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

78. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any TCE Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 68
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 10 [1 to 45] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 11 [1 to 48] | 0 [0 to 31] | 13 [1 to 53] | 0 [0 to 34] | 20 [3 to 56] | 0 [0 to 46] | 14 [1 to 58] | 0 [0 to 84]

79. Secondary Outcome: Percent of Responders: CD4+ T Cells With Any TCE Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 69
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0 [0 to 31] | 0 [0 to 31] | 13 [1 to 53] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

80. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Mem Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 70
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 10 [1 to 45] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 11 [1 to 48] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

81. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Mem Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 71
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0 [0 to 31] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

82. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Nuc Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 72
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0 [0 to 31] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 13 [1 to 53] | 0 [0 to 34] | 20 [3 to 56] | 0 [0 to 46] | 14 [1 to 58] | 0 [0 to 84]

83. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-Nuc Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 73
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 10 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0 [0 to 31] | 0 [0 to 31] | 13 [1 to 53] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

84. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-ORFa Stimulation Expressing IFNg and/or IL-2 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 74
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 9 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0 [0 to 31] | 0 [0 to 34] | 0 [0 to 37] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

85. Secondary Outcome: Percent of Responders: CD4+ T Cells With G-ORFa Stimulation Expressing IL-4 or IL-5 or IL-13 and CD154 for Groups 5, 6, 9, 10, 11, 13, 14 and 15
Description: as for outcome 75
Time Frame: Day 1 Pre-Vaccination, Day 15 Post Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of responders
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
percent of responders
  Day 1 Pre-Vaccination: number analyzed (Participants) | 10 | 9 | 8 | 8 | 10 | 6 | 7 | 2
  Day 1 Pre-Vaccination | 0 [0 to 31] | 0 [0 to 34] | 13 [1 to 53] | 0 [0 to 37] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]
  Day 15 Post-Vaccination: number analyzed (Participants) | 9 | 10 | 8 | 9 | 10 | 6 | 7 | 2
  Day 15 Post-Vaccination | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 37] | 0 [0 to 34] | 0 [0 to 31] | 0 [0 to 46] | 0 [0 to 41] | 0 [0 to 84]

86. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPs Spanning Membrane Frame for Groups 1 and 3A
Description: Mean spot forming units per million of the 15mer OLPs Spanning Membrane Frame as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 51.250 [-409.350 to 511.850]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 37.500 [-248.390 to 323.390]

87. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPa Spanning Nucleocapsid Frame for Groups 1 and 3A
Description: Mean spot forming units per million of the 15mer OLPa Spanning Nucleocapsid Frame as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 18.125 [8.180 to 28.070] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 42.500 [-32.796 to 117.796] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

88. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPs Spanning Open Reading Frame 3a for Groups 1 and 3A
Description: Mean spot forming units per million of the 15mer OLPs spanning Open Reading Frame 3a as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 16.875 [10.908 to 22.842] | 18.333 [3.991 to 32.676]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 29.375 [12.381 to 46.369] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 17.500 [9.544 to 25.456] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 21.667 [-7.018 to 50.351] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

89. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 1st of 4 OLP Pools for Groups 1 and 3A
Description: Mean spot forming units per million of the Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 17.500 [9.544 to 25.456] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 61.250 [36.407 to 86.093] | 29.167 [-31.788 to 90.121]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 120.000 [48.174 to 191.826] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 76.250 [19.571 to 132.929] | 37.500 [-248.390 to 323.390]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 257.500 [-342.980 to 857.980] | 230.000 [-2184.179 to 2644.179]

90. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 2nd of 4 OLP Pools for Groups 1 and 3A
Description: Mean spot forming units per million of the Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 131.875 [-119.329 to 383.079] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 250.625 [-187.616 to 688.866] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 140.625 [-41.568 to 322.818] | 25.000 [-102.062 to 152.062]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 525.833 [-912.305 to 1963.972] | 90.000 [-862.965 to 1042.965]

91. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 3rd of 4 OLP Pools for Groups 1 and 3A
Description: Mean spot forming units per million of the Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 18.333 [3.991 to 32.676]
  Day 29 Post Vaccination 1 | 60.625 [12.407 to 108,843] | 26.667 [-23.531 to 76.864]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 123.750 [74.224 to 173.276] | 19.167 [1.239 to 37.094]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 74.375 [22.775 to 125.975] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 241.667 [-291.170 to 774.503] | 166.250 [-1755.563 to 2088.063]

92. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 4th of 4 OLP Pools for Groups 1 and 3A
Description: Mean spot forming units per million of the Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 20.625 [10.163 to 31.087] | 17.500 [6.743 to 28.257]
  Day 29 Post Vaccination 1 | 16.875 [10.908 to 22.842] | 20.000 [-1.513 to 41.513]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 36.875 [9.052 to 64.698] | 27.500 [-11.284 to 66.284]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 49.375 [-19.326 to 118.076] | 28.750 [-145.960 to 203.460]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 75.833 [-67.723 to 219.389] | 177.500 [-1791.962 to 2146.962]

93. Secondary Outcome: Mean Spot Forming Units Per Million of the S1 for Groups 1 and 3A
Description: Mean spot forming units per million of the S1 as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 189.375 [-64.772 to 443.522] | 29.167 [-31.788 to 90.121]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 370.625 [-9.557 to 750.807] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 216.875 [68.016 to 365.734] | 55.000 [-453.248 to 563.248]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 775.000 [-858.462 to 2408.462] | 312.500 [-3149.941 to 3774.941]

94. Secondary Outcome: Mean Spot Forming Units Per Million of the S2 for Groups 1 and 3A
Description: Mean spot forming units per million of the S2 as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 60.625 [12.407 to 108.843] | 36.667 [-56.557 to 129.891]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 156.875 [82.923 to 230.827] | 25.000 [-18.027 to 68.027]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 120.000 [8.472 to 231.528] | 28.750 [-145.960 to 203.460]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 317.500 [-355.886 to 990.886] | 332.500 [-3701.720 to 4366.720]

95. Secondary Outcome: Mean Spot Forming Units Per Million of the Spike for Groups 1 and 3A
Description: Mean spot forming units per million of the Spike as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 250.000 [-52.175 to 552.175] | 55.833 [-119.858 to 231.525]
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 527.500 [109.835 to 945.165] | 25.000 [-18.027 to 68.027]
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 336.875 [194.760 to 478.990] | 76.250 [-702.005 to 854.505]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 1092.500 [-594.520 to 2779.520] | 637.500 [-6954.457 to 8229.457]

96. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLP (Overlapping Peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a for Groups 1 and 3A
Description: Mean spot forming units per million of the 15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a as measured by ELISpot
Time Frame: as for outcome 18
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 4 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1 (29 Days Post Vaccination 2) | 26.250 [5.579 to 46.921] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 4 | 2
  Day 209 Post Vaccination 1 (181 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 51.250 [-409.350 to 511.850]
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2): number analyzed (Participants) | 3 | 2
  Day 394 Post Vaccination 1 (366 Days Post Vaccination 2) | 54.167 [-69.157 to 177.491] | 37.500 [-248.390 to 323.390]

97. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPs Spanning Membrane Frame for Groups 3B and 4
Description: Mean spot forming units per million of the 15mer OLPs Spanning Membrane Frame as measured by ELISpot
Time Frame: Day 1 Pre-Vaccination 1, Day 29 Post Vaccination 1, Day 57 Post vaccination 1, Day 85 Post Vaccination 1, Day 99 Post Vaccination 1, Day 113 Post Vaccination 1, Day 169 Post Vaccination 1, Day 265 Post Vaccination 1
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 16.250 [13.037 to 19.463] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 16.250 [13.037 to 19.463] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 18.500 [8.782 to 28.218] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

98. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPa Spanning Nucleocapsid Frame for Groups 3B and 4
Description: Mean spot forming units per million of the 15mer OLPa Spanning Nucleocapsid Frame as measured by ELISpot
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 2
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 24.500 [-1.876 to 50.876] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

99. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPs Spanning Open Reading Frame 3a for Groups 3B and 4
Description: Mean spot forming units per million of the 15mer OLPs spanning Open Reading Frame 3a as measured by ELISpot
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 28.333 [-0.005 to 56.671] | 19.167 [1.239 to 37.094]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 37.917 [-16.015 to 91.848] | 27.500 [-7.078 to 62.078]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 40.000 [-29.155 to 109.155] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 18.750 [6.816 to 30.684] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 21.875 [-0.004 to 43.754] | 17.500 [6.743 to 28.257]
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 19.375 [11.174 to 27.576] | 23.333 [-12.522 to 59.189]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 17.083 [11.728 to 22.439] | 24.167 [-15.274 to 63.608]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 2
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

100. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 1st of 4 OLP Pools for Groups 3B and 4
Description: as for outcome 89
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 29.167 [8.134 to 50.199] | 20.000 [-1.513 to 41.513]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 34.167 [-4.057 to 72.391] | 24.167 [2.357 to 45.977]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 25.833 [-2.171 to 53.837] | 43.750 [-321.553 to 409.053]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 31.875 [-1.625 to 65.375] | 35.833 [-9.944 to 81.610]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 22.500 [8.342 to 36.658] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 33.125 [-1.153 to 67.403] | 17.500 [6.743 to 28.257]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 28.333 [-2.248 to 58.914] | 28.333 [-29.035 to 85.702]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 33.500 [14.927 to 52.073] | 328.333 [-688.521 to 1345.188]

101. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 2nd of 4 OLP Pools for Groups 3B and 4
Description: as for outcome 90
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 28.750 [2.318 to 55.182] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 17.500 [6.743 to 28.257]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 21.250 [1.360 to 41.140] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 16.875 [10.908 to 22.842] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 30.000 [0.504 to 59.496] | 72.500 [-174.903 to 319.903]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 304.500 [-478.516 to 1087.516] | 83.333 [-99.248 to 265.915]

102. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 3rd of 4 OLP Pools for Groups 3B and 4
Description: as for outcome 91
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 32.500 [-8.750 to 73.750] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 21.667 [6.038 to 37.296] | 20.000 [-43.531 to 83.531]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 20.000 [10.256 to 29.744] | 25.000 [0.159 to 49.841]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 31.250 [-2.739 to 65.239] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 21.875 [-0.004 to 43.754] | 22.500 [6.069 to 38.931]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 32.917 [-5.621 to 71.455] | 17.500 [6.743 to 28.257]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 85.000 [-51.935 to 221.935] | 74.167 [-110.306 to 258.639]

103. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 4th of 4 OLP Pools for Groups 3B and 4
Description: as for outcome 92
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 23.750 [11.699 to 35.801] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 19.167 [1.239 to 37.094] | 20.000 [-43.531 to 83.531]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 17.500 [9.544 to 25.456] | 21.667 [-7.018 to 50.351]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 17.500 [9.544 to 25.456] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 17.500 [9.544 to 25.456] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 17.500 [11.074 to 23.926] | 24.167 [-15.274 to 63.608]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 23.000 [5.523 to 40.477] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

104. Secondary Outcome: Mean Spot Forming Units Per Million of the S1 for Groups 3B and 4
Description: Mean spot forming units per million of the S1 as measured by ELISpot
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 27.917 [6.129 to 49.705] | 20.000 [-1.513 to 41.513]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 49.167 [-21.264 to 119.598] | 20.833 [-4.265 to 45.932]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 22.500 [-9.770 to 54.770] | 43.750 [-321.553 to 409.053]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 26.875 [-10.917 to 64.667] | 35.833 [-9.944 to 81.610]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 25.625 [5.504 to 45.746] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 33.125 [-1.153 to 67.403] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 44.583 [-5.097 to 94.263] | 90.833 [-235.451 to 417.118]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 324.500 [-469.444 to 1118.444] | 404.167 [-637.661 to 1445.994]

105. Secondary Outcome: Mean Spot Forming Units Per Million of the S2 for Groups 3B and 4
Description: Mean spot forming units per million of the S2 as measured by ELISpot
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 41.250 [-17.690 to 100.190] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 33.333 [-45.549 to 112.215]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 31.250 [-2.739 to 65.239] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 21.875 [-0.004 to 43.754] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 35.417 [-17.066 to 87.899] | 24.167 [-15.274 to 63.608]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 90.500 [-75.948 to 256.948] | 74.167 [-110.306 to 258.639]

106. Secondary Outcome: Mean Spot Forming Units Per Million of the Spike for Groups 3B and 4
Description: Mean spot forming units per million of the Spike as measured by ELISpot
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 27.917 [6.129 to 49.705] | 20.000 [-1.513 to 41.513]
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 77.917 [-57.135 to 212.968] | 20.833 [-4.265 to 45.932]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 22.500 [-9.770 to 54.770] | 43.750 [-321.553 to 409.053]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 26.875 [-10.917 to 64.667] | 59.167 [-76.090 to 194.423]
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 45.625 [2.734 to 88.516] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 40.000 [11.498 to 68.502] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 67.500 [-35.737 to 170.737] | 105.000 [-282.239 to 492.239]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 3
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 406.000 [-375.313 to 1187.313] | 473.333 [-616.760 to 1563.427]

107. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLP (Overlapping Peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a for Groups 3B and 4
Description: as for outcome 96
Time Frame: as for outcome 97
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 7 | 3
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 1 Pre-Vaccination 1 | 26.250 [-2.669 to 55.169] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post Vaccination 1: number analyzed (Participants) | 6 | 3
  Day 29 Post Vaccination 1 | 36.250 [-18.375 to 90.875] | 24.167 [-15.274 to 63.608]
  Day 57 Post vaccination 1: number analyzed (Participants) | 3 | 2
  Day 57 Post vaccination 1 | 40.000 [-29.155 to 109.155] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 4 | 3
  Day 85 Post Vaccination 1 | 18.750 [6.816 to 30.684] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 99 Post Vaccination 1 (15 Days Post Vaccination 2) | 21.875 [-0.004 to 43.754] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2): number analyzed (Participants) | 4 | 3
  Day 113 Post Vaccination 1 (29 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 23.333 [-12.522 to 59.189]
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2): number analyzed (Participants) | 6 | 3
  Day 169 Post Vaccination 1 (85 Days Post Vaccination 2) | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 24.167 [-15.274 to 63.608]
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2): number analyzed (Participants) | 5 | 2
  Day 265 Post Vaccination 1 (181 Days Post Vaccination 2) | 31.000 [-13.423 to 75.423] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal.

108. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPs Spanning Membrane Frame for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Mean spot forming units per million of the 15mer OLPs Spanning Membrane Frame as measured by ELISpot.
Time Frame: Day 1 Pre-Vaccination 1, Day 15 Post Vaccination 1, Day 29 Post vaccination 1, Day 85 Post Vaccination 1, Day 181 Post Vaccination 1
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 9 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 22.143 [12.295 to 31.991] | 17.778 [13.433 to 22.122] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 16.111 [13.549 to 18.673] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 21.944 [14.964 to 28.925] | 16.750 [12.791 to 20.709] | 18.438 [10.309 to 26.566] | 17.000 [13.984 to 20.016] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 18.93 [11.88 to 25.97] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 19.688 [11.445 to 27.930] | 18.889 [12.294 to 25.484] | 17.188 [12.015 to 22.360] | 16.000 [13.738 to 18.262] | 17.500 [11.735 to 23.265] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 17.813 [13.147 to 22.478] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 17.813 [13.423 to 22.202] | 20.250 [13.326 to 27.174] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 17.500 [13.657 to 21.343] | 22.813 [10.706 to 34.919] | 15.938 [13.721 to 18.154] | 30.750 [-4.879 to 66.379] | 16.111 [13.549 to 18.673] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

109. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPa Spanning Nucleocapsid Frame for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Mean spot forming units per million of the 15mer OLPa Spanning Nucleocapsid Frame as measured by ELISpot.
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 9 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 36.071 [10.573 to 61.570] | 35.556 [15.156 to 55.956] | 17.813 [11.162 to 24.463] | 17.778 [11.372 to 24.183] | 25.278 [1.577 to 48.978] | 16.79 [12.42 to 21.16] | 25.71 [-0.50 to 51.93] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal.
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 19.167 [12.373 to 25.961] | 25.500 [14.776 to 36.224] | 77.188 [-59.033 to 213.408] | 19.000 [9.951 to 28.049] | 17.500 [11.735 to 23.265] | 20.36 [11.87 to 28.84] | 28.93 [3.47 to 54.39] | 206.25 [-2223.81 to 2636.31]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 23.125 [16.732 to 29.518] | 28.333 [11.498 to 45.169] | 55.625 [-31.348 to 142.598] | 19.000 [9.951 to 28.049] | 18.611 [10.284 to 26.938] | 22.50 [10.64 to 34.36] | 45.00 [-4.47 to 94.47] | 666.25 [-7608.67 to 8941.17]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 25.938 [10.622 to 41.253] | 32.000 [11.284 to 52.716] | 64.375 [-29.772 to 158.522] | 21.500 [6.796 to 36.204] | 21.944 [5.931 to 37.958] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 28.75 [-15.01 to 72.51] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 51.111 [-12.798 to 115.020] | 34.688 [15.356 to 54.019] | 43.125 [3.113 to 83.137] | 36.750 [4.338 to 69.162] | 21.389 [6.656 to 36.122] | 17.50 [6.74 to 28.26] | 54.38 [-60.57 to 169.32] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

110. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLPs Spanning Open Reading Frame 3a for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Mean spot forming units per million of the 15mer OLPs spanning Open Reading Frame 3a as measured by ELISpot.
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 9 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 42.500 [-7.269 to 92.269] | 28.611 [1.433 to 55.790] | 20.938 [9.882 to 31.993] | 15.000 [NA to NA] — 95% CI was not estimable because all values were equal. | 22.500 [7.247 to 37.753] | 19.64 [10.95 to 28.34] | 17.14 [13.76 to 20.53] | 31.25 [-175.23 to 237.73]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 9 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 46.667 [21.101 to 72.233] | 18.889 [12.294 to 25.484] | 31.250 [6.369 to 56.131] | 19.250 [11.339 to 27.161] | 20.556 [11.605 to 29.506] | 26.07 [6.55 to 45.59] | 26.79 [0.88 to 52.69] | 70.00 [-628.84 to 768.84]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 44.063 [27.307 to 60.818] | 31.944 [2.116 to 61.773] | 42.188 [9.512 to 74.863] | 21.250 [7.112 to 35.388] | 28.056 [8.136 to 47.975] | 29.29 [10.95 to 47.62] | 27.50 [-0.95 to 55.95] | 157.50 [-1557.84 to 1872.84]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 26.250 [14.166 to 38.334] | 22.750 [8.088 to 37.412] | 37.813 [13.530 to 62.095] | 22.000 [13.536 to 30.464] | 24.167 [6.925 to 41.408] | 17.50 [9.54 to 25.46] | 20.63 [2.72 to 38.53] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 30.278 [4.885 to 55.671] | 34.688 [14.472 to 54.903] | 23.750 [10.159 to 37.341] | 24.000 [3.641 to 44.359] | 19.722 [8.833 to 30.612] | 18.33 [3.99 to 32.68] | 18.13 [8.18 to 28.07] | 22.50 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

111. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 1st of 4 OLP Pools for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: as for outcome 89
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 193.214 [0.407 to 386.022] | 148.000 [58.422 to 237.578] | 109.688 [-26.303 to 245.678] | 56.389 [23.804 to 88.974] | 137.500 [-119.160 to 394.160] | 118.21 [38.91 to 197.52] | 197.50 [-70.02 to 465.02] | 208.75 [-2157.78 to 2575.28]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 160.278 [80.381 to 240.174] | 130.000 [51.905 to 208.095] | 137.813 [43.595 to 232.030] | 117.000 [7.183 to 226.817] | 117.500 [-31.708 to 266.708] | 132.50 [21.40 to 243.60] | 437.86 [-118.32 to 994.03] | 827.50 [-8416.26 to 10071.26]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 153.438 [109.271 to 197.604] | 151.000 [46.413 to 255.587] | 163.750 [-3.987 to 331.487] | 146.000 [-51.075 to 343.075] | 117.222 [-36.870 to 271.314] | 140.71 [51.48 to 229.95] | 431.25 [-119.11 to 981.61] | 1157.50 [-12025.19 to 14340.19]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 118.438 [69.359 to 167.516] | 157.000 [85.242 to 228.758] | 170.313 [45.436 to 295.189] | 117.750 [-6.487 to 241.987] | 105.278 [-79.354 to 289.909] | 73.75 [17.26 to 130.24] | 412.50 [-403.44 to 1228.44] | 40.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 201.389 [-8.577 to 411.355] | 195.938 [-36.806 to 428.681] | 112.500 [49.204 to 175.796] | 210.750 [-110.210 to 531.710] | 95.833 [-50.419 to 242.086] | 82.50 [-20.86 to 185.86] | 415.00 [-327.27 to 1157.27] | 45.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

112. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 2nd of 4 OLP Pools for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: as for outcome 90
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 151.429 [51.197 to 251.660] | 188.250 [83.786 to 292.714] | 118.438 [-12.291 to 249.166] | 61.389 [30.536 to 92.242] | 124.167 [-26.541 to 274.874] | 108.57 [25.71 to 191.43] | 58.57 [-3.85 to 121.00] | 576.25 [-6555.11 to 7707.61]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 143.056 [107.417 to 178.694] | 143.500 [47.780 to 239.220] | 116.563 [38.201 to 194.924] | 104.500 [24.918 to 184.082] | 124.167 [19.753 to 228.580] | 127.14 [33.69 to 220.60] | 87.86 [-9.64 to 185.35] | 1006.25 [-11048.76 to 13061.26]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 146.875 [93.545 to 200.205] | 183.889 [61.342 to 306.436] | 150.625 [-17.364 to 318.614] | 115.000 [35.154 to 194.846] | 131.667 [-2.010 to 265.344] | 139.64 [41.41 to 237.88] | 93.75 [3.97 to 183.53] | 1360.00 [-15634.55 to 18354.55]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 101.563 [68.744 to 134.381] | 158.750 [65.547 to 251.953] | 155.938 [14.868 to 297.007] | 101.750 [33.880 to 169.620] | 116.667 [-10.516 to 243.849] | 95.00 [-9.50 to 199.50] | 83.13 [-79.26 to 245.51] | 25.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 143.611 [81.260 to 205.963] | 486.875 [-264.121 to 1237.871] | 125.313 [43.335 to 207.290] | 166.750 [-61.320 to 394.820] | 79.167 [-4.321 to 162.654] | 122.50 [-144.11 to 389.11] | 81.25 [-17.08 to 179.58] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

113. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 3rd of 4 OLP Pools for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: as for outcome 91
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 193.929 [35.278 to 352.579] | 225.250 [59.864 to 390.636] | 103.438 [-8.943 to 215.818] | 101.111 [28.786 to 173.437] | 180.556 [-150.518 to 511.630] | 182.14 [45.45 to 318.83] | 126.43 [-42.46 to 295.31] | 65.00 [-570.31 to 700.31]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 159.444 [86.720 to 232.169] | 155.500 [66.695 to 244.305] | 128.438 [41.837 to 215.038] | 132.750 [30.697 to 234.803] | 134.772 [-48.040 to 317.484] | 256.43 [111.50 to 401.36] | 225.71 [-66.22 to 517.65] | 206.25 [-1906.16 to 2318.66]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 151.250 [56.652 to 245.848] | 173.611 [61.415 to 285.807] | 128.750 [7.697 to 249.803] | 126.750 [21.176 to 232.324] | 137.500 [-72.220 to 347.220] | 269.29 [113.82 to 424.75] | 245.42 [-117.80 to 608.64] | 451.25 [-4742.41 to 5644.91]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 130.625 [52.648 to 208.602] | 199.000 [69.122 to 328.878] | 139.063 [40.074 to 238.051] | 119.000 [41.022 to 196.978] | 135.833 [-106.303 to 377.969] | 156.88 [32.33 to 281.42] | 336.88 [-596.26 to 1270.01] | 30.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 241.667 [36.450 to 446.883] | 215.000 [4.700 to 425.300] | 94.688 [46.565 to 142.810] | 233.000 [-136.739 to 602.739] | 109.444 [-47.953 to 266.842] | 198.33 [-20.47 to 417.14] | 217.50 [-274.50 to 709.50] | 22.50 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

114. Secondary Outcome: Mean Spot Forming Units Per Million of the Consensus Spike (Wuhan-1) Whole Protein, 4th of 4 OLP Pools for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: as for outcome 92
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 83.929 [-7.196 to 175.053] | 91.500 [19.770 to 163.230] | 44.688 [18.334 to 71.041] | 45.556 [8.110 to 83.001] | 53.333 [-7.306 to 113.973] | 91.79 [35.19 to 148.38] | 47.50 [5.12 to 89.88] | 31.25 [15.37 to 47.13]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 84.167 [43.857 to 124.476] | 83.750 [22.768 to 144.732] | 53.125 [12.601 to 93.649] | 72.750 [28.344 to 117.156] | 64.444 [32.120 to 96.769] | 108.93 [60.49 to 157.37] | 48.93 [9.38 to 88.48] | 91.25 [-496.41 to 678.91]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 81.250 [45.361 to 117.139] | 91.944 [28.531 to 155.358] | 67.500 [23.616 to 111.384] | 80.500 [23.441 to 137.559] | 58.333 [16.177 to 100.490] | 121.43 [70.18 to 172.68] | 50.42 [19.98 to 80.85] | 78.75 [-254.79 to 412.29]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 56.563 [28.994 to 84.131] | 71.250 [15.035 to 127.465] | 61.875 [29.733 to 94.017] | 67.750 [21.134 to 114.366] | 79.722 [-6.595 to 166.039] | 69.38 [42.91 to 95.84] | 47.50 [-48.14 to 143.14] | 25.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 72.778 [17.687 to 127.868] | 157.500 [-65.975 to 380.975] | 42.813 [18.325 to 67.300] | 77.250 [7.861 to 146.639] | 51.944 [12.918 to 90.971] | 80.83 [-48.30 to 209.96] | 32.50 [6.72 to 58.28] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

115. Secondary Outcome: Mean Spot Forming Units Per Million of the S1 for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Mean spot forming units per million of the S1 as measured by ELISpot.
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 344.643 [73.157 to 616.128] | 334.000 [152.907 to 515.093] | 224.375 [-43.540 to 492.290] | 110.833 [47.142 to 174.524] | 247.778 [-157.638 to 653.194] | 223.57 [72.86 to 374.28] | 246.79 [-66.71 to 560.28] | 773.75 [-8867.08 to 10414.58]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 303.333 [204.591 to 402.075] | 268.500 [102.559 to 434.441] | 249.375 [76.426 to 422.324] | 213.500 [25.430 to 401.570] | 243.722 [10.040 to 459.405] | 259.64 [83.16 to 436.12] | 516.43 [-140.55 to 1173.41] | 1833.75 [-19465.03 to 23132.53]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 300.313 [215.957 to 384.668] | 348.333 [119.531 to 577.135] | 306.875 [-29.828 to 643.578] | 254.250 [-12.757 to 521.257] | 237.500 [-35.436 to 510.436] | 276.43 [99.66 to 453.20] | 520.83 [-103.49 to 1145.16] | 2506.25 [-27813.93 to 32826.43]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 218.125 [147.869 to 288.381] | 313.250 [171.078 to 455.422] | 322.500 [58.245 to 586.755] | 212.750 [21.941 to 403.559] | 209.444 [-90.550 to 509.439] | 165.00 [5.84 to 324.16] | 488.13 [-490.54 to 1466.79] | 40.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 345.000 [84.088 to 605.912] | 674.375 [-213.067 to 1561.817] | 230.313 [86.993 to 373.632] | 371.000 [-179.486 to 921.486] | 160.556 [-72.268 to 393.379] | 196.67 [-198.77 to 592.10] | 486.25 [-361.95 to 1334.45] | 45.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

116. Secondary Outcome: Mean Spot Forming Units Per Million of the S2 for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Mean spot forming units per million of the S2 as measured by ELISpot.
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 271.786 [28.289 to 515.282] | 308.750 [76.000 to 541.500] | 138.438 [0.228 to 276.647] | 136.667 [23.349 to 249.984] | 223.889 [-169.836 to 617.613] | 273.93 [86.23 to 461.62] | 164.64 [-50.29 to 379.58] | 88.75 [-657.74 to 835.24]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 238.611 [138.564 to 338.659] | 233.750 [90.039 to 377.461] | 174.688 [54.237 to 295.138] | 191.500 [40.265 to 342.735] | 190.278 [-18.107 to 398.663] | 365.36 [190.84 to 539.87] | 263.57 [-67.56 to 594.70] | 297.50 [-2402.57 to 2997.57]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 232.500 [111.741 to 353.259] | 262.222 [100.318 to 424.126] | 185.938 [20.814 to 351.061] | 202.750 [42.937 to 362.563] | 185.556 [-66.879 to 437.990] | 390.71 [200.45 to 580.98] | 289.58 [-99.30 to 678.46] | 530.00 [-4997.20 to 6057.20]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 183.438 [81.132 to 285.743] | 262.750 [98.821 to 426.679] | 190.313 [55.127 to 325.498] | 178.750 [56.888 to 300.612] | 203.056 [-126.882 to 532.993] | 226.25 [93.89 to 358.61] | 368.75 [-676.45 to 1413.95] | 30.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 311.111 [50.230 to 571.992] | 365.938 [-65.269 to 797.144] | 130.313 [54.283 to 206.342] | 303.500 [-135.520 to 742.520] | 149.722 [-47.484 to 346.929] | 279.17 [-59.87 to 618.20] | 238.75 [-289.24 to 766.74] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

117. Secondary Outcome: Mean Spot Forming Units Per Million of the Spike for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: Mean spot forming units per million of the Spike as measured by ELISpot.
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 10 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 616.429 [104.946 to 1127.911] | 641.250 [239.386 to 1043.114] | 360.938 [-38.143 to 760.018] | 245.833 [74.320 to 417.347] | 466.667 [-331.690 to 1265.023] | 497.50 [163.29 to 831.71] | 407.14 [-65.93 to 880.22] | 855.00 [-9627.62 to 11337.62]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 10 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 541.944 [361.956 to 721.933] | 500.750 [198.369 to 803.131] | 424.063 [139.388 to 708.737] | 399.000 [61.306 to 736.694] | 423.333 [-1.042 to 847.708] | 625.00 [284.20 to 965.80] | 775.71 [-196.03 to 1747.46] | 2131.25 [-21867.59 to 26130.09]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 532.813 [345.095 to 720.530] | 610.556 [236.649 to 984.462] | 492.813 [-5.871 to 991.496] | 452.500 [33.223 to 871.777] | 418.056 [-104.235 to 940.346] | 667.14 [313.09 to 1021.20] | 807.92 [-142.87 to 1758.71] | 3036.25 [-32811.13 to 38883.63]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 401.563 [246.202 to 556.923] | 576.000 [288.467 to 863.533] | 510.938 [117.787 to 904.088] | 390.000 [86.109 to 693.891] | 405.833 [-220.889 to 1032.556] | 391.25 [100.83 to 681.67] | 849.38 [-1148.74 to 2847.49] | 70.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 656.111 [138.931 to 1173.291] | 1038.438 [-163.839 to 2240.714] | 360.625 [147.341 to 573.909] | 670.000 [-320.087 to 1660.087] | 305.278 [-124.952 to 735.507] | 475.83 [-257.94 to 1209.61] | 717.50 [-597.31 to 2014.31] | 45.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

118. Secondary Outcome: Mean Spot Forming Units Per Million of the 15mer OLP (Overlapping Peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a for Groups 5, 6, 9, 10, 11, 13, 14, and 15
Description: as for outcome 96
Time Frame: as for outcome 108
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: SFU/million cells
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 7 | 7 | 2
SFU/million cells
  Day 1 Pre-Vaccination 1: number analyzed (Participants) | 7 | 9 | 8 | 9 | 9 | 7 | 7 | 2
  Day 1 Pre-Vaccination 1 | 72.143 [-9.586 to 153.871] | 48.611 [15.353 to 81.869] | 22.500 [10.416 to 34.584] | 17.778 [11.372 to 24.183] | 33.611 [-9.306 to 76.528] | 18.57 [9.83 to 27.31] | 25.71 [-0.50 to 51.93] | 31.25 [-175.23 to 237.73]
  Day 15 Post Vaccination 1: number analyzed (Participants) | 9 | 9 | 8 | 10 | 9 | 7 | 7 | 2
  Day 15 Post Vaccination 1 | 62.222 [28.614 to 95.830] | 33.056 [17.362 to 48.749] | 97.813 [-65.874 to 261.499] | 22.500 [11.158 to 33.842] | 24.722 [9.276 to 40.169] | 38.57 [-2.83 to 79.97] | 38.57 [5.69 to 71.46] | 268.75 [-2955.45 to 3492.95]
  Day 29 Post vaccination 1: number analyzed (Participants) | 8 | 9 | 8 | 10 | 9 | 7 | 6 | 2
  Day 29 Post vaccination 1 | 57.500 [33.801 to 81.199] | 49.444 [9.356 to 89.533] | 89.688 [-21.495 to 200.870] | 25.250 [9.333 to 41.167] | 37.500 [3.097 to 71.903] | 31.07 [10.57 to 51.57] | 58.75 [-20.82 to 138.32] | 812.50 [-9320.70 to 10945.70]
  Day 85 Post Vaccination 1: number analyzed (Participants) | 8 | 10 | 8 | 10 | 9 | 4 | 4 | 1
  Day 85 Post Vaccination 1 | 39.063 [17.546 to 60.579] | 37.500 [14.259 to 60.741] | 90.938 [-25.018 to 206.893] | 37.500 [5.464 to 69.536] | 32.778 [-4.092 to 69.647] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 34.38 [-7.01 to 75.76] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.
  Day 181 Post Vaccination 1: number analyzed (Participants) | 9 | 8 | 8 | 10 | 9 | 3 | 4 | 1
  Day 181 Post Vaccination 1 | 68.611 [-24.303 to 161.525] | 72.500 [14.289 to 130.711] | 53.750 [12.173 to 95.327] | 63.750 [-30.692 to 158.192] | 27.778 [-1.688 to 57.243] | 15.00 [NA to NA] — 95% CI was not estimable because all values were equal. | 51.88 [-65.48 to 169.23] | 15.00 [NA to NA] — 95% CI was not estimable because only one participant was analyzed at this time point.

119. Secondary Outcome: Mean T-cells Expressing IL-2 in pg/mL for Groups 1 and 3A at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-2 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: The mITT population includes all enrolled participants who received at least one dose vaccine and contributed both pre- and at least one post vaccination venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. The Group 1 arm consists of 3 participants as 1 participant did not have any data reported for this outcome.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 17.651 [-26.698 to 62.000] | 5.290 [-6.633 to 17.213]
  15mer OLPa Spanning Nucleocapsid Frame | 10.427 [-8.247 to 29.100] | 16.898 [-28.172 to 61.967]
  15mer OLPs spanning Open Reading Frame 3a | 21.312 [-44.758 to 87.382] | 17.151 [-7.616 to 41.917]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 109.721 [-25.788 to 245.230] | 24.202 [-41.440 to 89.845]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 99.148 [-120.489 to 318.785] | 18.059 [-16.388 to 52.506]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 87.137 [-79.954 to 254.228] | 35.403 [-58.048 to 128.854]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 31.072 [-31.944 to 94.089] | 17.899 [-14.819 to 50.617]
  S1 | 208.869 [-139.777 to 557.515] | 42.261 [-56.755 to 141.278]
  S2 | 118.209 [-108.211 to 344.629] | 53.302 [-71.694 to 178.299]
  Spike | 327.078 [-246.801 to 900.957] | 95.564 [-128.256 to 319.383]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 49.390 [-74.127 to 172.907] | 39.339 [-20.521 to 99.198]

120. Secondary Outcome: Mean T-cells Expressing IL-4 in pg/mL for Groups 1 and 3A at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-4 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 119
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.084 [-0.113 to 0.281] | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPa Spanning Nucleocapsid Frame | 0.128 [-0.079 to 0.335] | 0.082 [-0.107 to 0.271]
  15mer OLPs spanning Open Reading Frame 3a | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.053 [-0.013 to 0.119]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 0.492 [-1.018 to 2.002] | 0.131 [-0.270 to 0.532]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 0.176 [-0.187 to 0.539] | 0.120 [-0.081 to 0.321]
  S1 | 0.492 [-1.018 to 2.002] | 0.131 [-0.270 to 0.532]
  S2 | 0.176 [-0.187 to 0.539] | 0.120 [-0.081 to 0.321]
  Spike | 0.656 [-1.223 to 2.534] | 0.226 [-0.441 to 0.862]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 0.174 [0.100 to 0.248] | 0.097 [-0.069 to 0.264]

121. Secondary Outcome: Mean T-cells Expressing IL-10 in pg/mL for Groups 1 and 3A at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-10 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 119
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.085 [0.022 to 0.148] | 1.852 [-5.255 to 8.985]
  15mer OLPa Spanning Nucleocapsid Frame | 0.761 [-0.046 to 1.569] | 5.044 [-16.357 to 26.445]
  15mer OLPs spanning Open Reading Frame 3a | 0.387 [-0.803 to 1.576] | 4.479 [-13.349 to 22.307]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 1.837 [0.022 to 3.651] | 10.422 [-32.497 to 53.340]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 1.557 [-1.150 to 4.263] | 8.160 [-24.018 to 40.338]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 0.740 [-0.685 to 2.164] | 8.377 [-27.366 to 44.121]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 0.486 [-0.408 to 1.379] | 5.005 [-15.816 to 25.827]
  S1 | 3.393 [-0.379 to 7.166] | 18.558 [-56.585 to 93.701]
  S2 | 1.225 [-1.045 to 3.495] | 13.336 [-43.328 to 70.000]
  Spike | 4.618 [-1.152 to 10.388] | 31.871 [-99.986 to 163.728]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 1.125 [-0.392 to 2.641] | 11.304 [-35.175 to 57.783]

122. Secondary Outcome: Mean T-cells Expressing IL-13 in pg/mL for Groups 1 and 3A at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-13 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 119
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 5.252 [-5.918 to 16.422] | 4.728 [-2.353 to 11.790]
  15mer OLPa Spanning Nucleocapsid Frame | 2.597 [-1.907 to 7.101] | 2.279 [-0.856 to 5.413]
  15mer OLPs spanning Open Reading Frame 3a | 2.124 [-0.346 to 4.595] | 2.156 [-0.451 to 4.763]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 3.361 [2.020 to 4.701] | 2.156 [-0.451 to 4.763]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 6.043 [-2.915 to 15.000] | 5.175 [-4.396 to 14.746]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 2.342 [0.606 to 4.078] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 3.736 [-3.185 to 10.657] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  S1 | 7.645 [-0.619 to 15.909] | 6.298 [-7.810 to 20.405]
  S2 | 3.324 [-4.310 to 10.959] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Spike | 9.936 [8.286 to 11.586] | 6.298 [-7.810 to 20.405]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 7.390 [-5.848 to 20.628] | 7.095 [-8.863 to 23.054]

123. Secondary Outcome: Mean T-cells Expressing TNF-alpha in pg/mL for Groups 1 and 3A at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing TNF-alpha in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 119
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 8.845 [-10.475 to 28.166] | 12.990 [-32.235 to 58.215]
  15mer OLPa Spanning Nucleocapsid Frame | 6.784 [-2.998 to 16.565] | 27.390 [-78.121 to 132.900]
  15mer OLPs spanning Open Reading Frame 3a | 6.100 [-10.727 to 22.927] | 18.547 [-52.294 to 89.388]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 17.145 [0.386 to 33.904] | 72.302 [-215.814 to 360.418]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 18.845 [-29.049 to 66.739] | 35.237 [-99.111 to 169.585]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 9.712 [-6.629 to 26.052] | 44.250 [-134.450 to 222.950]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 7.229 [-5.170 to 19.628] | 27.882 [-82.377 to 138.140]
  S1 | 35.990 [-28.290 to 100.270] | 107.539 [-314.880 to 529.958]
  S2 | 16.941 [-11.798 to 45.679] | 72.131 [-216.817 to 361.080]
  Spike | 52.931 [-39.561 to 145.422] | 179.671 [-531.688 to 891.029]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 21.729 [-24.130 to 67.588] | 58.926 [-162.607 to 280.460]

124. Secondary Outcome: Mean T-cells Expressing IL-2 in pg/mL for Groups 3B and 4 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-2 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: The mITT population includes all enrolled participants who received at least one dose vaccine and contributed both pre- and at least one post vaccination venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. The Group 3B arm consists of 2 participants as 5 participants did not have any data reported for this outcome. The Group 4 arm consists of 2 participants as 1 participant did not have any data reported for this outcome.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 2 | 2
pg/mL
  15mer OLPs Spanning Membrane Frame | 5.246 [-9.591 to 20.084] | 11.715 [-3.949 to 27.378]
  15mer OLPa Spanning Nucleocapsid Frame | 956.979 [-11025.246 to 12939.203] | 10.155 [0.651 to 19.659]
  15mer OLPs spanning Open Reading Frame 3a | 32.492 [-46.226 to 111.210] | 9.801 [-18.521 to 38.123]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 41.112 [-28.985 to 111.209] | 25.725 [9.874 to 41.575]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 6.923 [-32.972 to 46.817] | 12.611 [-11.500 to 36.721]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 17.987 [-15.408 to 51.382] | 21.148 [-109.252 to 151.549]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 16.322 [-0.333 to 32.976] | 16.493 [4.263 to 28.723]
  S1 | 48.035 [-61.957 to 158.026] | 38.335 [30.076 to 46.594]
  S2 | 34.309 [-15.741 to 84.358] | 37.641 [-80.530 to 155.812]
  Spike | 82.343 [-77.698 to 242.384] | 75.976 [-33.936 to 185.888]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 994.717 [-11081.063 to 13070.497] | 31.671 [9.508 to 53.834]

125. Secondary Outcome: Mean T-cells Expressing IL-4 in pg/mL for Groups 3B and 4 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-4 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 124
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 2 | 2
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.299 [-0.864 to 1.462]
  15mer OLPa Spanning Nucleocapsid Frame | 36.585 [-425.445 to 498.614] | 0.063 [-0.255 to 0.381]
  15mer OLPs spanning Open Reading Frame 3a | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.186 [-1.260 to 1.631]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.126 [-0.995 to 1.248]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.601 [0.182 to 1.020]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 0.082 [-0.480 to 0.644] | 0.075 [-0.389 to 0.538]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.260 [-0.868 to 1.387]
  S1 | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.708 [-1.074 to 2.490]
  S2 | 0.082 [-0.480 to 0.644] | 0.315 [-0.107 to 0.738]
  Spike | 0.082 [-0.480 to 0.644] | 1.024 [-1.181 to 3.228]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 36.585 [-425.445 to 498.614] | 0.493 [-2.014 to 2.999]

126. Secondary Outcome: Mean T-cells Expressing IL-10 in pg/mL for Groups 3B and 4 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-10 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 124
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 2 | 2
pg/mL
  15mer OLPs Spanning Membrane Frame | 12.384 [-122.197 to 146.965] | 0.569 [0.486 to 0.651]
  15mer OLPa Spanning Nucleocapsid Frame | 329.048 [-3803.325 to 4461.420] | 0.499 [-2.315 to 3.313]
  15mer OLPs spanning Open Reading Frame 3a | 26.108 [-263.975 to 316.190] | 0.657 [-2.202 to 3.515]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 22.599 [-47.914 to 93.112] | 1.934 [-4.778 to 8.646]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 15.392 [-121.365 to 152.149] | 1.158 [-2.534 to 4.849]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 30.663 [-291.084 to 352.410] | 1.144 [-0.819 to 3.107]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 11.987 [-100.279 to 124.252] | 0.522 [-0.339 to 1.383]
  S1 | 37.991 [-169.279 to 245.261] | 3.091 [-7.312 to 13.494]
  S2 | 42.650 [-391.363 to 476.662] | 1.666 [0.563 to 2.768]
  Spike | 80.641 [-560.642 to 721.923] | 4.757 [-6.748 to 16.262]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 367.540 [-4189.496 to 4924.575] | 1.724 [-4.032 to 7.480]

127. Secondary Outcome: Mean T-cells Expressing IL-13 in pg/mL for Groups 3B and 4 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-13 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 124
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 2 | 2
pg/mL
  15mer OLPs Spanning Membrane Frame | 3.460 [-20.806 to 27.725] | 9.699 [-11.108 to 30.505]
  15mer OLPa Spanning Nucleocapsid Frame | 193.308 [-2218.133 to 2604.748] | 4.304 [0.825 to 7.782]
  15mer OLPs spanning Open Reading Frame 3a | 3.897 [-9.442 to 17.235] | 10.186 [1.085 to 19.287]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 3.953 [-26.577 to 34.483] | 10.869 [-7.695 to 29.432]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 4.015 [-27.309 to 35.339] | 8.758 [-34.291 to 51.806]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 4.833 [-36.881 to 46.547] | 6.204 [-18.376 to 30.784]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 4.609 [-34.259 to 43.477] | 10.498 [-14.232 to 35.227]
  S1 | 7.193 [-64.508 to 78.894] | 19.626 [-41.986 to 81.238]
  S2 | 8.667 [-81.763 to 99.097] | 16.702 [-32.608 to 66.011]
  Spike | 15.085 [-156.893 to 187.063] | 36.328 [-74.594 to 147.250]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 198.466 [-2147.437 to 2544.368] | 24.188 [-2.241 to 50.617]

128. Secondary Outcome: Mean T-cells Expressing TNF-alpha in pg/mL for Groups 3B and 4 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing TNF-alpha in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 124
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 2 | 2
pg/mL
  15mer OLPs Spanning Membrane Frame | 128.731 [-1278.592 to 1536.055] | 3.194 [-14.585 to 20.973]
  15mer OLPa Spanning Nucleocapsid Frame | 1861.230 [-21502.562 to 25225.021] | 3.744 [-11.380 to 18.867]
  15mer OLPs spanning Open Reading Frame 3a | 300.416 [-3311.513 to 3912.345] | 3.433 [1.766 to 5.101]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 167.163 [-1370.904 to 1705.230] | 10.697 [-9.744 to 31.138]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 145.340 [-1474.361 to 1765.041] | 5.505 [-1.083 to 12.093]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 290.681 [-3172.723 to 3754.084] | 6.443 [-7.658 to 20.543]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 123.765 [-1132.231 to 1379.760] | 6.927 [-39.381 to 53.235]
  S1 | 312.503 [-2845.265 to 3470.271] | 16.202 [-10.828 to 43.231]
  S2 | 414.445 [-4304.954 to 5133.844] | 13.370 [-47.039 to 73.778]
  Spike | 726.948 [-7150.219 to 8604.115] | 29.572 [-57.866 to 117.009]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 2290.337 [-26092.667 to 30673.421] | 10.371 [-20.864 to 41.606]

129. Secondary Outcome: Mean T-cells Expressing IL-2 in pg/mL for Groups 3B and 4 at Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Description: Mean T-cells Expressing IL-2 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Population: The mITT population includes all enrolled participants who received at least one dose vaccine and contributed both pre- and at least one post vaccination venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. The Group 3B arm consists of 3 participants as 4 participants did not have any data reported for this outcome.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 13.754 [-15.746 to 43.255] | 18.749 [-24.999 to 62.498]
  15mer OLPa Spanning Nucleocapsid Frame | 5.648 [-4.696 to 15.993] | 11.485 [5.361 to 17.609]
  15mer OLPs spanning Open Reading Frame 3a | 15.310 [-9.570 to 40.190] | 12.042 [6.083 to 18.000]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 24.703 [-9.748 to 59.153] | 31.098 [8.617 to 53.579]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 24.621 [-25.412 to 74.654] | 20.411 [-10.602 to 51.424]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 25.392 [3.517 to 47.267] | 24.891 [9.533 to 40.249]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 32.809 [7.250 to 58.367] | 31.035 [-25.135 to 87.205]
  S1 | 49.324 [-28.085 to 126.732] | 51.509 [12.617 to 890.401]
  S2 | 58.201 [39.136 to 77.265] | 55.926 [6.785 to 105.067]
  Spike | 107.524 [18.334 to 196.714] | 107.435 [85.905 to 128.965]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 34.713 [-9.368 to 78.793] | 42.267 [4.842 to 79.709]

130. Secondary Outcome: Mean T-cells Expressing IL-4 in pg/mL for Groups 3B and 4 at Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Description: Mean T-cells Expressing IL-4 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 129
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPa Spanning Nucleocapsid Frame | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPs spanning Open Reading Frame 3a | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 0.047 [0.007 to 0.087] | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  S1 | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  S2 | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Spike | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.

131. Secondary Outcome: Mean T-cells Expressing IL-10 in pg/mL for Groups 3B and 4 at Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Description: Mean T-cells Expressing IL-10 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 129
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.808 [-1.071 to 2.687] | 0.161 [-0.037 to 0.359]
  15mer OLPa Spanning Nucleocapsid Frame | 1.208 [-1.299 to 3.715] | 0.156 [-0.215 to 0.528]
  15mer OLPs spanning Open Reading Frame 3a | 1.072 [-1.499 to 3.643] | 0.070 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 6.466 [-6.123 to 19.054] | 2.167 [-0.821 to 5.156]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 3.250 [-6.541 to 13.041] | 0.391 [-0.509 to 1.290]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 2.050 [-3.687 to 7.787] | 1.064 [-0.516 to 2.644]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 1.538 [-2.160 to 5.236] | 0.341 [-0.123 to 0.806]
  S1 | 9.715 [-12.623 to 32.053] | 2.534 [-1.035 to 6.104]
  S2 | 3.565 [-5.910 to 13.040] | 1.361 [-0.812 to 3.534]
  Spike | 13.257 [-18.587 to 45.101] | 3.895 [-1.769 to 9.559]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 3.042 [-4.085 to 10.168] | 0.271 [-0.346 to 0.887]

132. Secondary Outcome: Mean T-cells Expressing IL-13 in pg/mL for Groups 3B and 4 at Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Description: Mean T-cells Expressing IL-13 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 129
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 3.796 [-5.868 to 13.461] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPa Spanning Nucleocapsid Frame | 4.089 [-1.868 to 10.046] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPs spanning Open Reading Frame 3a | 3.404 [-1.897 to 8.704] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal. | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 5.534 [-3.050 to 14.117] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 1.990 [0.097 to 3.882] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 3.485 [-0.679 to 7.649] | 1.880 [0.459 to 3.302]
  S1 | 5.534 [-3.050 to 14.117] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  S2 | 3.485 [-0.679 to 7.649] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Spike | 8.502 [-6.458 to 23.462] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 8.764 [-12.848 to 30.376] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.

133. Secondary Outcome: Mean T-cells Expressing TNF-alpha in pg/mL for Groups 3B and 4 at Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Description: Mean T-cells Expressing TNF-alpha in pg/mL as measured by MSD cytokine assay
Time Frame: Day 113 Post Vaccination 1 (29 Days Post Vaccination 2)
Population: as for outcome 129
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 5.400 [2.225 to 8.575] | 3.213 [1.238 to 5.188]
  15mer OLPa Spanning Nucleocapsid Frame | 7.971 [-0.802 to 16.744] | 4.853 [-4.970 to 14.677]
  15mer OLPs spanning Open Reading Frame 3a | 6.162 [3.692 to 8.633] | 1.989 [-1.134 to 5.113]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 18.952 [8.464 to 29.440] | 13.546 [1.295 to 25.796]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 8.549 [2.027 to 15.072] | 5.384 [-1.534 to 12.302]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 9.284 [5.387 to 13.182] | 7.804 [-2.993 to 18.601]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 7.486 [2.208 to 12.763] | 5.214 [2.196 to 8.232]
  S1 | 27.501 [23.446 to 31.556] | 18.930 [-0.212 to 38.071]
  S2 | 16.770 [7.628 to 25.911] | 13.018 [2.007 to 24.029]
  Spike | 44.271 [38.797 to 49.745] | 31.948 [1.796 to 62.099]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 19.533 [8.308 to 30.759] | 10.056 [-4.766 to 24.877]

134. Secondary Outcome: Mean T-cells Expressing IL-2 in pg/mL for Groups 5 and 6 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-2 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: The mITT population includes all enrolled participants who received at least one dose vaccine and contributed both pre- and at least one post vaccination venous blood sample for the corresponding immunogenicity endpoint testing and for which valid results were reported. The Group 5 and 6 arms consist of 3 participants as 7 participants in each arm did not have any data reported for this outcome.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 15.533 [-7.734 to 38.800] | 15.847 [-15.260 to 46.954]
  15mer OLPa Spanning Nucleocapsid Frame | 16.116 [-35.309 to 67.540] | 19.297 [9.430 to 29.164]
  15mer OLPs spanning Open Reading Frame 3a | 26.168 [-21.150 to 73.487] | 15.559 [-12.381 to 43.500]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 129.978 [-26.833 to 280.788] | 732.268 [-1781.612 to 3246.148]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 87.681 [40.903 to 134.459] | 755.178 [-1720.997 to 3231.353]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 91.627 [41.985 to 141.269] | 727.250 [-1796.013 to 3250.513]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 51.847 [-6.682 to 110.376] | 689.798 [-1913.803 to 3293.398]
  S1 | 214.659 [15.434 to 413.883] | 1487.446 [-3499.827 to 6474.719]
  S2 | 143.474 [130.879 to 156.068] | 1417.047 [-3709.505 to 6543.599]
  Spike | 358.132 [152.738 to 563.527] | 2904.493 [-7203.839 to 13012.825]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 57.817 [-54.718 to 170.351] | 50.703 [2.394 to 99.013]

135. Secondary Outcome: Mean T-cells Expressing IL-4 in pg/mL for Groups 5 and 6 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-4 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 134
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.047 [0.007 to 0.087]
  15mer OLPa Spanning Nucleocapsid Frame | 0.109 [-0.129 to 0.347] | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPs spanning Open Reading Frame 3a | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 0.059 [-0.031 to 0.149] | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 0.076 [-0.007 to 0.158] | 0.052 [-0.009 to 0.113]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.056 [-0.023 to 0.135]
  S1 | 0.097 [0.080 to 0.114] | 0.052 [-0.009 to 0.113]
  S2 | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal. | 0.056 [-0.023 to 0.135]
  Spike | 0.097 [0.080 to 0.114] | 0.071 [-0.001 to 0.142]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 0.098 [-0.160 to 0.356] | 0.038 [NA to NA] — 95% CI was not estimable because all values were equal.

136. Secondary Outcome: Mean T-cells Expressing IL-10 in pg/mL for Groups 5 and 6 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-10 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 134
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 0.438 [-1.145 to 2.021] | 1.264 [-1.181 to 3.709]
  15mer OLPa Spanning Nucleocapsid Frame | 1.124 [-1.271 to 3.518] | 2.151 [-2.251 to 6.552]
  15mer OLPs spanning Open Reading Frame 3a | 0.778 [-1.270 to 2.826] | 2.972 [-3.942 to 9.887]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 6.628 [-4.934 to 18.190] | 21.391 [-15.156 to 57.939]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 1.533 [-1.047 to 4.112] | 5.901 [-4.033 to 15.834]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 1.541 [-2.614 to 5.695] | 5.602 [-3.234 to 14.438]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 1.021 [-1.755 to 3.796] | 3.856 [-0.787 to 8.500]
  S1 | 8.160 [-5.656 to 21.976] | 27.292 [-18.886 to 73.469]
  S2 | 2.561 [-4.259 to 9.382] | 9.458 [-2.042 to 20.959]
  Spike | 10.722 [-9.787 to 31.230] | 36.750 [-20.243 to 93.743]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 2.269 [-3.824 to 8.363] | 6.348 [-7.359 to 20.055]

137. Secondary Outcome: Mean T-cells Expressing IL-13 in pg/mL for Groups 5 and 6 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing IL-13 in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 134
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 3.205 [-0.359 to 6.768] | 3.558 [-2.315 to 9.431]
  15mer OLPa Spanning Nucleocapsid Frame | 2.692 [-2.223 to 7.607] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  15mer OLPs spanning Open Reading Frame 3a | 2.622 [0.315 to 4.928] | 1.909 [0.365 to 3.453]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 2.935 [-3.024 to 8.893] | 1.550 [NA to NA] — 95% CI was not estimable because all values were equal.
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 2.716 [0.125 to 5.307] | 3.376 [-0.623 to 7.375]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 2.072 [-0.175 to 4.320] | 1.990 [0.097 to 3.882]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 1.938 [0.270 to 3.605] | 2.757 [-2.437 to 7.952]
  S1 | 3.605 [-1.556 to 8.766] | 3.376 [-0.623 to 7.375]
  S2 | 2.072 [-0.175 to 4.320] | 2.757 [-2.437 to 7.952]
  Spike | 4.644 [-4.684 to 13.972] | 5.100 [-4.414 to 14.613]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 6.452 [0.977 to 11.927] | 3.088 [-3.529 to 9.705]

138. Secondary Outcome: Mean T-cells Expressing TNF-alpha in pg/mL for Groups 5 and 6 at Day 29 Post Vaccination 1
Description: Mean T-cells Expressing TNF-alpha in pg/mL as measured by MSD cytokine assay
Time Frame: Day 29 Post Vaccination 1
Population: as for outcome 134
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6
Number analyzed (Participants) | 3 | 3
pg/mL
  15mer OLPs Spanning Membrane Frame | 7.161 [-1.168 to 15.490] | 11.752 [-9.290 to 32.793]
  15mer OLPa Spanning Nucleocapsid Frame | 10.909 [-0.194 to 22.012] | 20.224 [-16.584 to 57.032]
  15mer OLPs spanning Open Reading Frame 3a | 7.423 [-5.791 to 20.636] | 16.296 [-12.389 to 44.982]
  Consensus Spike (Wuhan-1) whole protein, 1st of 4 OLP pools | 30.201 [8.447 to 51.954] | 209.438 [-72.520 to 491.395]
  Consensus Spike (Wuhan-1) whole protein, 2nd of 4 OLP pools | 12.700 [-1.047 to 26.446] | 96.215 [-107.586 to 300.016]
  Consensus Spike (Wuhan-1) whole protein, 3rd of 4 OLP pools | 14.317 [3.558 to 25.076] | 68.809 [-58.408 to 196.027]
  Consensus Spike (Wuhan-1) whole protein, 4th of 4 OLP pools | 10.754 [-4.612 to 26.120] | 71.193 [-84.607 to 226.993]
  S1 | 42.900 [7.621 to 78.180] | 305.653 [-149.208 to 760.514]
  S2 | 25.071 [-0.986 to 51.128] | 140.002 [-142.724 to 422.728]
  Spike | 67.971 [6.724 to 129.219] | 445.655 [-252.526 to 1143.836]
  15mer OLP (overlapping peptides) Spanning Membrane, Nucleocapsid, and Open Reading Frame 3a | 25.493 [-6.663 to 57.649] | 48.272 [-37.362 to 133.905]

ADVERSE EVENTS:
Time Frame: Solicited AEs (i.e., reactogenicity) were collected from the time of each study vaccination through 7 days post each study vaccination. Unsolicited AEs of all severities were reported from the time of study product administration through 28 days post each vaccination.
Description: After 28 days post last vaccination through the end of study, only SAEs, AESIs (including PIMMCs, NOCMCs, and MAAEs), and AEs leading to withdrawal from the study were reported. All participants were followed through 12 months after their last study vaccination.
Arm/Group | Stage 1 (Naïve) Group 1 | Stage 1 (Naïve) Group 3A | Stage 1 (Naïve) Group 3B | Stage 1 (Naïve) Group 4 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/7 | 0/3 | 0/10 | 0/10 | 0/8 | 0/10 | 0/10 | 0/7 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/7 | 0/3 | 0/10 | 0/10 | 0/8 | 0/10 | 0/10 | 0/7 | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 7/7 | 3/3 | 10/10 | 10/10 | 8/8 | 10/10 | 10/10 | 7/7 | 7/7 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 (Naïve) Group 1 (N=4) | Stage 1 (Naïve) Group 3A (N=3) | Stage 1 (Naïve) Group 3B (N=7) | Stage 1 (Naïve) Group 4 (N=3) | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 5 (N=10) | Stage 2 (SAM-S-TCE Boosts After EUA/Licensed mRNA COVID-19 Vaccines) Group 6 (N=10) | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 9 (N=8) | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 10A,B (N=10) | Stage 2 (SAM-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 11A,B (N=10) | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 13 (N=7) | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 14 (N=7) | Stage 2 (ChAd-S-TCE Boosts After Approved/Licensed mRNA COVID-19 Vaccines) Group 15 (N=2)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (5) | 5 (6) | 1 (2) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (6) | 3 (5) | 7 (11) | 3 (5) | 5 (5) | 7 (7) | 3 (3) | 5 (5) | 7 (7) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 4 (7) | 2 (3) | 7 (12) | 3 (6) | 9 (9) | 8 (8) | 7 (7) | 9 (9) | 8 (8) | 3 (3) | 4 (4) | 2 (2)
Injection site pain (General disorders) | 4 (6) | 2 (3) | 7 (12) | 3 (5) | 9 (9) | 10 (10) | 7 (7) | 6 (6) | 10 (10) | 1 (1) | 4 (4) | 2 (2)
Malaise (General disorders) | 4 (6) | 3 (5) | 7 (13) | 3 (6) | 5 (5) | 5 (5) | 6 (6) | 5 (5) | 8 (8) | 2 (2) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 3 (4) | 7 (10) | 3 (5) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Vaccination site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site induration (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 4 (8) | 3 (4) | 7 (13) | 3 (6) | 10 (10) | 8 (8) | 5 (5) | 8 (8) | 9 (9) | 1 (1) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 0 (0) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (5) | 6 (8) | 3 (5) | 5 (5) | 5 (5) | 6 (6) | 6 (6) | 8 (8) | 1 (1) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 3 (5) | 3 (5) | 6 (11) | 3 (6) | 6 (6) | 8 (8) | 4 (4) | 8 (8) | 7 (7) | 1 (1) | 4 (4) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 5 (5) | 2 (2) | 5 (5) | 1 (1) | 5 (6) | 4 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT04776317/Prot_002.pdf
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04776317/SAP_000.pdf
  • Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04776317/ICF_001.pdf